Statistical Analysis Plan: J2G-OX-JZJG

A Single-Dose, Randomized, Double-Blind, Placebo- and Positive-Controlled, 4-Way Crossover Study to Evaluate the Effect of LOXO-292 on the QTc Interval in Healthy Adult Subjects

NCT05630274

Approval Date: 24-Jul-2019



- **16.1.9 Documentation of Statistical Methods**
- 16.1.9.1 Statistical Analysis Plan

## Statistical Analysis Plan

A Single-Dose, Randomized, Double-Blind, Placebo- and Positive-Controlled, 4-Way Crossover Study to Evaluate the Effect of LOXO-292 on the QTc Interval in Healthy Adult Subjects

> Protocol No: LOXO-RET-18032 Final Protocol Date: 03 April 2019 Protocol Clarification Letter: 18 April 2019 Compound Name: LOXO-292

> > Celerion Project CA25494 Final Version 1.0 Date: 28 June 2019

Loxo Oncology, Inc. 701 Gateway Boulevard, Suite 420 South San Francisco, California 94080, USA

Celerion
621 Rose Street
Lincoln, Nebraska 68502, USA
And
100 Alexis-Nihon Boulevard, Suite 360,
Montreal, QC H4M 2N8, Canada

## Statistical Analysis Plan Signature Page

Compound Name: LOXO-292

Protocol: LOXO-RET-18032

Study Title: A Single-Dose, Randomized, Double-Blind, Placebo- and Positive-Controlled, 4-Way Crossover Study to Evaluate the Effect of LOXO-292 on the QTc Interval in Healthy Adult Subjects

Issue Date: 28 June 2019

| Signatu | PPD | Date: 05/4/2019 |
|---|---|---|
| | Director, Biostatistics, Data Management<br>Celerion, PPD USA | t and Biometrics |
| Signature | PPD | Date: 04 - JUL - 2019 |
| | PPD Clinical Pharmata Management and Biometrics Celerion, PPD Canada | nacology and Pharmacometrics, |
| Signatur | PPD | 11-Jul-19 17:41:16 PDT<br>Date: |
| | | California, USA |

## **Table of Contents**

| 1.? | INTF | ODUCTION | 5 |
|---|---|---|---|
| 2.? | OBJI | ECTIVES AND ENDPOINTS | 5 |
| | 2.12 | Objectives | 5 |
| | 2.2? | Endpoints | 6 |
| 3.? | STU | DY DESIGN | 6 |
| 4.2 | ANA | LYSIS POPULATIONS | 7 |
| | | Analysis Populations | |
| | | Preliminary Data and Interim Analysis | |
| <b>5</b> .? | TRE | ATMENT DESCRIPTIONS | 8 |
| 6.2 | PHA | RMACOKINETIC ANALYSIS | 9 |
| | 6.12 | Measurements and Collection Schedule | 9 |
| | | Bioanalytical Method | |
| | | 6.2.12 LOXO-292 | 9 |
| | | 6.2.2 Moxifloxacin | 10 |
| | 6.32 | Investigational Product and PK Analyte Information | 10 |
| | | 6.3.12 LOXO-292 | 10 |
| | | 6.3.2 Moxifloxacin | 10 |
| | 6.42 | Pharmacokinetic Concentrations | 10 |
| | 6.52 | Noncompartmental Pharmacokinetic Analysis and Parameter Calculation for LOXO-292 and Moxifloxacin | 10 |
| | 6.62 | Data Summarization and Presentation | |
| 7.2 | SAFI | ETY | 13 |
| | | Subject Discontinuation | |
| | 7.2 | Demographics | |
| | 7.32 | Adverse Events | 13 |
| | 7.42 | Clinical Laboratory Tests (Serum Chemistry, Hematology, Coagulation, and Urinalysis) | 15 |
| | 7.52 | Vital Signs (Blood Pressure, Pulse Rate, Respiration Rate, and Temperature) | 17 |
| | 7.62 | Safety ECG (Heart Rate, PR, QRS, QT, and QTcF [QT with Fridericia correction]) | |
| | <b>7 7</b> ? | Concomitant Medications | |
| | | Physical Examination | |
| 8.2 | | MARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS | |
| 9.? | SUM | MARY TABLES AND FIGURES | 18 |
| | 9.12 | In-text Summary Tables and Figures | 19 |
| | 9.27 | Section 14 Summary Tables and Figures | 19 |

## Loxo Oncology, Inc. LOXO-292, LOXO-RET-18032 Celerion, Clinical Study Report No. CA25494

| 9.32 Section 16 Data Listings | 22 |
|-------------------------------|----|
| 10. TABLE AND FIGURE SHELLS | |
| 10.12 In-text Table Shells | |
| 10.22 Figures Shells | |
| 10.32 Post-text Table Shells | |
| 11.DLISTING SHELLS | 57 |

#### 1. INTRODUCTION

The following statistical analysis plan (SAP) provides the framework for the summarization of the data from study LOXO-RET-18032 which will be analyzed by Celerion. The SAP may change due to unforeseen circumstances. Any changes made from the planned analysis within the protocol or after the locking of the database will be documented in the clinical study report (CSR). The section referred to as Table Shells within this SAP describes the traceability of the tables, figures, and listings (TFLs) back to the data. Note that the header for this page will be the one used for the main body of the CSR.

Any additional analyses not addressed within this SAP and/or driven by the data, or requested by Loxo Oncology, Inc., will be considered out of scope and will be described in the CSR as needed.

## 2. OBJECTIVES AND ENDPOINTS

## 2.1 Objectives

Celerion will only assess the 3rd and 4th secondary objectives which are bolded below. All other objectives will be assessed by ERT (eResearchTechnology, Inc.) in a separate SAP and study report.

#### **Primary:**

To evaluate the effects of therapeutic and supratherapeutic exposure of LOXO-292 on the heart rate-corrected (QTc) interval by assessing concentration-QT (C-QT) relationship using exposure-response modelling.

#### Secondary:

To assess the effect of therapeutic and supratherapeutic exposure of LOXO-292 on other electrocardiogram (ECG) parameters.

To demonstrate sensitivity of this QTc assay using moxifloxacin as a positive control in healthy adult subjects.

To evaluate the pharmacokinetics (PK) of therapeutic and supratherapeutic doses of LOXO-292 in healthy adult subjects.

To evaluate the safety and tolerability of therapeutic and supratherapeutic doses of LOXO-292 dose in healthy adult subjects.



#### 2.2 Endpoints

The cardiodynamic endpoints will be addressed will be addressed by ERT.

#### **Pharmacokinetics:**

The following PK parameters will be calculated for LOXO-292 and moxifloxacin: AUC0-t, AUC0-inf, AUC%extrap, Cmax, Tmax, Kel, and t½.

## Safety:

Safety endpoints will include 12-lead ECGs, physical examinations, vital signs, clinical laboratory tests, and adverse events (AEs).

## 3. STUDY DESIGN

This is a single-dose, randomized, double-blind (except for the use of moxifloxacin), placebo- and positive-controlled, 4-way crossover study.

Thirty-two (32), healthy, adult male and female (women of non-childbearing potential only) subjects will be enrolled.

Screening of subjects will occur within 28 days prior to the first dosing.

On Day 1, subjects will be randomized to 1 of 4 treatment sequences.

On Day 1 of each period, subjects will receive one of two single oral dose levels of LOXO-292, a single oral dose of moxifloxacin, or a single oral dose of LOXO-292 matching placebo on one occasion, according to a randomization scheme. Cardiodynamic samples will be collected predose and for up to 24 hours postdose. PK samples will be collected predose and for up to 24 hours postdose for moxifloxacin and up to 240 hours postdose for LOXO-292, as per treatment received.

There will be a washout period of 10 days between dosing in each period.

Safety and tolerability will be assessed through End of Treatment (EOT) or Early Termination (ET) by monitoring AEs, performing physical examinations and clinical laboratory tests, measuring vital signs, and recording ECGs.

Subjects who do not complete the study treatments will not be replaced.

Subjects will be housed through EOT or ET beginning in Period 1, Day -1, at the time indicated by the clinical research unit (CRU), until after completion of study procedures in Period 4, Day 11 (EOT) or ET study procedures.

The CRU will contact all subjects who received at least one dose of study drug (including subjects who terminated the study early [ET]) at the End of Study (EOS) by a follow up (FU) phone call. The EOS/FU phone call will be performed  $7 \pm 2$  days after the EOT visit or ET visit to determine if any SAE or study drug related AE has occurred since the EOT or ET visit.

#### 4. ANALYSIS POPULATIONS

#### 4.1 Analysis Populations

## **Safety Population**

All subjects who received at least one dose of either of the study drugs will be included in the safety evaluations.

## Pharmacokinetic Population

Samples from all subjects will be assayed even if the subjects do not complete the study. All subjects who comply sufficiently with the protocol and display an evaluable PK profile (e.g., exposure to treatment, availability of measurements and absence of major protocol violations) will be included in the statistical analyses.

Data for each subject will be included in the summary statistics and statistical comparisons of PK parameters with the exceptions described as follows:

- Data from subjects who experience emesis at or before 2 times median Tmax for the given treatment during the PK sampling period time course of the study for LOXO-292 or moxifloxacin may be excluded from the summary statistics for the given treatment and from the statistical comparison of PK parameters.
- Data from subjects who significantly violate a protocol inclusion or exclusion criterion, deviate significantly from the protocol, or have unavailable or incomplete data that may influence the PK analysis will be excluded from the PK Population.

Any subject or data excluded from the analysis will be identified, along with their reason for exclusion, in the CSR.

## 4.2 Preliminary Data and Interim Analysis

No interim analysis is planned for this study.

## 5. TREATMENT DESCRIPTIONS

LOXO-292 will be supplied as completed mg CC

LOXO-292 matching placebo will be supplied as CC

Moxifloxacin will be supplied as mg Avelox® (moxifloxacin hydrochloride) or generic equivalent cl.

Treatments are described as follows:

Treatment A: mg LOXO-292 (mg CCl m) and LOXO-292 matching placebo (mg mg matching placebo CCl m) administered at Hour 0 on Day 1.

Treatment B: mg LOXO-292 ( mg CC ) administered at Hour 0 on Day 1.

Treatment C: mg moxifloxacin (1 x CC mg CCI) administered at Hour 0 on Day 1.

Treatment D: LOXO-292 matching placebo (CCI m) mg matching placebo CCI administered at Hour 0 on Day 1.

Each treatment will be administered orally following a fast of at least 10 hours from food (not including water), with approximately 240 mL of water. Subjects will remain (not including water) for at least 4 hours postdose.

Subjects will be instructed not to crush, split, or chew the CCI or the CCI.

The pharmacy at the CRU will provide each dose in individual unit dose containers for each subject and for each study period.

**Table 5.1 Treatment Description** 

| Treatment | Short Description (text, figure legends, SAS output) | Description (listings footnotes, intext and post-text tables footnotes) |
|---|---|---|
| A | mg LOXO-292 | mg LOXO-292 ( mg mg mg loxO-292 matching placebo ( mg mg mg |

| В | mg LOXO-292 | mg LOXO-292 ( mg CC mg ) administered at Hour 0 on Day 1 |
|---|---|---|
| С | ccl mg moxifloxacin | mg moxifloxacin (1 x CCI mg CCI) administered at Hour 0 on Day 1 |
| D | LOXO-292 matching placebo | LOXO-292 matching placebo mg matching placebo CCI and a distribution of the control of the con |

#### 6. PHARMACOKINETIC ANALYSIS

#### 6.1 Measurements and Collection Schedule

PK samples will be collected predose and for up to 24 hours postdose for moxifloxacin and up to 240 hours postdose for LOXO-292.

Blood samples for PK assessment of LOXO-292 will be taken at the following time points for Treatments A, B, and D: at predose and 0.25, 0.5, 0.75, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, and 240 hours postdose.

Blood samples for PK assessment of moxifloxacin will be taken at the following time points for Treatment C: at predose and 0.25, 0.5, 0.75, 1.5, 2, 2.5, 3, 4, 7, 9, 12, and 24 hours postdose.

All concentration data will be included in the calculation of the individual PK parameters, the individual concentration-time plots (based on actual sample times), and in the mean concentration-time plots (based on nominal sample times). However, if there are any significant deviations from nominal sample times, some concentration data may be excluded from mean concentration-time plots and/or additional concentration-time plots of the mean data may be provided. All deviations and excluded data will be provided and discussed in the CSR.

## 6.2 Bioanalytical Method

## 6.2.1 LOXO-292

Plasma concentrations of LOXO-292 in Treatments A, B, and D will be determined using a liquid chromatography-tandem mass spectrometry (LC-MS/MS) method validated with respect to accuracy, precision, linearity, sensitivity, and specificity at

Alturas Analytics, Inc. (Moscow, Idaho, USA). The analytical range (lower limit of quantitation [LLOQ] – upper limit of quantitation [ULOQ]) for LOXO-292 in plasma is 1-1000 ng/mL. Samples that contain concentrations greater than 1000 ng/mL may be diluted up to 51-fold, if necessary, to be within the quantification range.

#### 6.2.2 Moxifloxacin

Plasma concentrations of moxifloxacin in Treatment C will be determined using a LC-MS/MS method validated with respect to accuracy, precision, linearity, sensitivity, and specificity at Alturas Analytics, Inc. (Moscow, Idaho, USA). The analytical range (LLOQ – ULOQ) for moxifloxacin in plasma is 25 – 25000 ng/mL.

## 6.3 Investigational Product and PK Analyte Information

#### 6.3.1 LOXO-292

LOXO-292 will be supplied as a simple blend with excipients containing of drug substance (freebase) in a hard gelatin capsule.

#### 6.3.2 Moxifloxacin

Moxifloxacin will be supplied as a **CCI** containing **CCI**mg drug substance.

#### 6.4 Pharmacokinetic Concentrations

Plasma concentrations of LOXO-292 and moxifloxacin as determined at the collection times and per the bioanalytical methods described in Section 6.1 and Section 6.2, respectively, will be used for the calculation of the plasma LOXO-292 and moxifloxacin PK parameters.

## 6.5 Noncompartmental Pharmacokinetic Analysis and Parameter Calculation for LOXO-292 and Moxifloxacin

The appropriate noncompartmental PK parameters will be calculated from the plasma LOXO-292 and moxifloxacin concentration-time data using Phoenix® WinNonLin® Version 7.0 or higher. Actual sample collection times will be used in the calculations of the PK parameters. The calculation of the actual time for LOXO-292 and moxifloxacin will be in respect to the administration time of the LOXO-292 and moxifloxacin dose, respectively. All PK parameters included in the protocol are listed in Table 6.1 below, and are defined as appropriate for study design.

Table 6.1. Noncompartmental Pharmacokinetic Parameters to be Calculated for LOXO-292 and Moxifloxacin

| Label to be<br>Used in the<br>Text, Tables<br>and Figures | Definition | Method of Determination |
|---|---|---|
| AUC0-t | Area under the concentration-time curve from time 0 to the time of the last observed non-zero concentration | Calculated using the Linear Trapezoidal with Linear Interpolation Method |
| AUC0-inf | Area under the concentration-time curve from time 0 extrapolated to infinity | Calculated as AUC0-t + (Clast/Kel) where Clast is the last observed/measured concentration |
| AUC%extrap | Percent of AUC0-inf extrapolated | Calculated as 1-(AUC0-t/AUC0-inf)*100 |
| Cmax | Maximum observed concentration | Taken directly from bioanalytical data |
| Tmax | The time to reach Cmax. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value | Taken from clinical database as the difference in the time of administration and the time of the blood draw which is associated with the Cmax. |
| Kel | Apparent terminal elimination rate constant; represents the fraction of drug eliminated per unit time | Calculated as the negative of the slope of a linear regression of the log(concentration)-time for all concentrations >LLOQ during the terminal elimination phase |
| t½ | Apparent first-order terminal elimination half-life | Calculated as 0.693/Kel |

PK parameters will not be calculated for subjects with fewer than 3 consecutive postdose time points with quantifiable concentrations. Subjects for whom there are insufficient data to calculate the PK parameters will be included in the concentration tables only and excluded from all statistical analysis.

For the calculation of the PK parameters and PK concentrations summary statistics, plasma concentrations below the limit of quantitation (BLQ) prior to the first quantifiable concentration of a PK profile will be set to 0 and plasma concentrations BLQ after the first quantifiable concentration of a PK profile will be treated as missing.

The Kel will be determined using linear regressions composed of least 3 data points. The Kel will not be assigned if 1) the terminal elimination phase is not apparent, 2) if Tmax is one of the 3 last data points, or 3) if the R<sup>2</sup> value is less than 0.75. In cases where the Kel interval is not assigned, the values of t½, AUC0-inf, and AUC%extrap are considered not calculable and will not be reported. Wherever the resulting t½ is more than half as long as the sampling interval, the Kel values and associated

parameters (t½, AUC0-inf, and AUC%extrap) may not be presented as judged appropriate and in accordance with Celerion SOPs.

#### 6.6 Data Summarization and Presentation

All LOXO-292 and moxifloxacin PK concentrations and PK parameters descriptive statistics will be generated using SAS® Version 9.3 or higher.

The plasma concentrations of LOXO-292 and moxifloxacin will be listed and summarized by treatment and time point for all subjects in the PK Population. Plasma concentrations of LOXO-292 and moxifloxacin will be presented with the same level of precision as received from the bioanalytical laboratory. Summary statistics, including sample size (n), arithmetic mean (Mean), standard deviation (SD), coefficient of variation (CV%), standard error of the mean (SEM), minimum, median, and maximum will be calculated for all nominal concentration time points. Excluded subjects will be included in the concentration listings, but will be excluded from the summary statistics and noted as such in the tables. All BLQ values will be presented as "BLQ" in the concentration listings and footnoted accordingly.

Mean and individual concentration-time profiles will be presented on linear and semilog scales. Linear mean plots will be presented with and without SD.

Plasma LOXO-292 and moxifloxacin PK parameters will be listed and summarized by treatment for all subjects in the PK Population. PK parameters will be reported to 3 significant figures for individual parameters, with the exception of Tmax and t½, which will be presented with 2 decimal places. Summary statistics (n, Mean, SD, CV%, SEM, minimum, median, maximum, geometric mean [Geom Mean] and geometric CV% [Geom CV%]) will be calculated for plasma LOXO-292 and moxifloxacin PK parameters. Excluded subjects will be listed in the PK parameter tables, but will be excluded from the summary statistics and noted as such in the tables.

The level of precision for each concentration and PK parameter statistic will be presented as follows:

- minimum/maximum in same precision as in bioanalytical data and parameter output,
- mean/median/Geom Mean in one more level of precision than minimum/maximum,
- SD/SEM in one more level of precision than mean/median/Geom Mean,
- n will be presented as an integer, and
- CV%/ Geom CV% will be presented to the nearest tenth.

No inferential statistics will be performed on PK concentrations or parameters.

#### 7. SAFETY

No inferential statistics are to be performed for the safety analysis.

All clinical safety and tolerability data will be listed by subject and assessment time points, including rechecks, unscheduled assessments, and early termination (ET), chronologically.

Continuous variables will be summarized using n, mean, SD, minimum, median, and maximum. Frequency counts will be reported for categorical data when appropriate.

The level of precision will be presented as follows: "n" as an integer, minimum/maximum in same precision as in the database, mean/median in one more precision level than minimum/maximum, and SD in one more precision level than mean/median.

Where individual data points are missing because of dropouts or other reasons, the data will be summarized based on reduced denominators.

When change from baseline is calculated, baseline is the last scheduled assessment before dosing, including rechecks and unscheduled assessments, whichever is later, unless otherwise specified in the sections below. Rechecks, unscheduled assessments and ET measurements taken after dosing will not be used in the summarization.

## 7.1 Subject Discontinuation

Subjects will be summarized by the number of subjects enrolled, completed, and discontinued from the study with discontinuation reasons by randomized treatment sequence and overall. Discontinuation data will be listed by-subject.

## 7.2 Demographics

Descriptive statistics will be calculated for continuous variables (age, weight, height, and body mass index) for randomized treatment sequence and study overall. Weight, height and body mass index are summarized at screening. Age will be derived from the date of birth to the date of first dosing at Period 1. Frequency counts will be provided for categorical variables (race, ethnicity, and sex) for overall. A by-subject listing will also be provided.

#### 7.3 Adverse Events

All AEs occurring during this clinical trial will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®), Version 22.0.

Each AE will be graded, by the clinical site, on the National Institution of Health's Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) 5-point severity scale (Grade 1, 2, 3, 4 and 5). Not all grades are appropriate for all AEs. Therefore, some AEs are listed within the CTCAE with fewer than 5 options for grade selection.

The following clinical descriptions of severity for each AE are based on the following general guideline [CTCAE Nov2017]:

Table 7.3: Adverse Event Severity Level and Description

| Grade | Description |
|---|---|
| Grade 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. |
| Grade 2 | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL)*. |
| Grade 3 | Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL**. |
| Grade 4 | Life-threatening consequences; urgent intervention indicated. |
| Grade 5 | Death related to AE. |

<sup>\*</sup> Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

Similarly, the causal relationship of the study drugs to the AE will be described as Related or Unrelated to study drugs LOXO-292 or moxifloxacin.

All AEs captured in the database will be listed in by-subject data listings including verbatim term, coded term, treatment group, severity grade, relationship to study drugs, and action; however, only treatment-emergent AEs (TEAEs) will be summarized.

A TEAE is defined as an undesirable event not present prior to medical treatment, or an already present event that worsens either in intensity or frequency following the treatment. Each TEAE will be attributed to a treatment based on Investigator (or

<sup>\*\*</sup> Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications and not bedridden.□

designee) judgment as well as on its onset date and time. An AE that occurs during the washout period between treatments will be considered treatment-emergent to the last treatment given. If an AE has a change in severity grade, the original AE will be given a resolution date and time of the time of severity grade increase or decrease and a new AE record will be initiated with the new severity grade, and the new AE record will use the resolved date/time of the previous record as the onset date/time. If an AE decreases in severity grade, the new AE record with less severity will be considered and counted as the same AE event of the previous record with worse severity under the same treatment group and period in the analysis. If the severity grade of an AE remains the same, the AE will be kept open through to resolution.

If the onset time of an AE is missing and the onset date is the same as the treatment dosing date, then the AE will be considered treatment-emergent in both the prior and current treatment. If the onset time of an AE is missing and the onset date does not fall on a dosing date, then the AE will be considered treatment-emergent for the last treatment administered. If the onset date of an AE is missing, then the AE will be considered treatment-emergent and attributed to the first treatment group on the study, unless the onset date is known to have occurred within or between specific treatment periods.

TEAEs will be tabulated by system organ class and preferred term. Summary tables will include the number of subjects reporting the AE and as a percent of the number of subjects dosed by treatment and overall. Tables will also be presented by severity grade and relationship to study drugs. If a subject experienced the same TEAE at more than once with different level of severity grade for a given treatment, only the most severe one will be counted. Similarly, if a subject experienced the same TEAE at more than once with different level of drug relationship for a given treatment, only the one most closely related to each study drug will be counted.

Should any serious adverse events (SAEs) occur during the study, the SAEs will be displayed in a table and a narrative included in the CSR.

## 7.4 Clinical Laboratory Tests (Serum Chemistry, Hematology, Coagulation, and Urinalysis)

All clinical laboratory test results will be presented in by-subject data listings, however, only serum chemistry, hematology, coagulation and urinalysis values will be summarized.

Hematology, coagulation, serum chemistry and urinalysis tests will be conducted at the following time points:

**Table 7.4 Lab Test Time Points** 

| Period | Period Day |
|--------|------------|
| Screen | |

| 1 | Day -1 (check-in) |
|---|---|
| 1-4 | Day 3, Day 6, Day 11 |
| End of | |
| Treatment/Early | |
| Termination | |
| Period Day 1 in Periods 2-4 is the same as Period Day 11 of the | |
| previous period. | |

Out-of-normal range (OOR) flags will be recorded as follows: high (H) and low (L) for numerical results and did-not-match (\*) for categorical results. If a value fails the reference range, it will automatically be compared to a computer clinically significant (CS) range suggested by the PI (Celerion SOP GSOP.10.1028). If the value falls within the computer CS range, it will be noted as "N" for not clinically significant. If the value fails (i.e., falls outside of the CS range) the computer CS range, it will be flagged with a "Y" which prompts the PI to determine how the OOR value should be followed using 4 Investigator flags: "N", not clinically significant, "R", requesting a recheck, "^", checking at the next scheduled visit, or "Y", clinically significant. To distinguish the PI flag from the CS range flags, the PI flags "N" and "Y" will be presented as "-" and "+" in the data listings, respectively. Additionally, the PI will provide a 4<sup>th</sup> flag when the 3<sup>rd</sup> flag indicates "R" or "^". This 4<sup>th</sup> flag is intended to capture final CS (+)/NCS (-) when the 3<sup>rd</sup> flag does not document significance. In addition, CTCAE, version 5.0 grading (found in NCI CTCAE guidance) will be applied to all out of range lab values deemed clinically significant by the Investigator (or designee) which are recorded as AEs.

Out-of-range values and corresponding recheck results will be listed. Results that are indicated as CS by the PI (in either PI flag) will be listed in the table. Out-of-range values laboratory value results which are indicated as CS by PI will be reported as AEs.

For all laboratory values that are numeric, descriptive statistics (n, mean, SD, minimum, median, and maximum) will be presented for each laboratory test by treatment and time point. Change from baseline will also be summarized. Postdose unscheduled events or rechecks will not be summarized. Similarly, ET results will not be included in summaries.

For each laboratory test, a shift table will be developed comparing the frequency of the results at baseline (above normal, normal, or below normal) to postdose results. For urinalysis tests, the categories are normal and outside normal.

Baseline is Day -1 of Period 1 and Day 11 of previous period for Periods 2, 3, 4 and is the last non-missing predose measurement prior to dosing, including rechecks and unscheduled assessments. Day 11 measurement of Periods 1, 2, 3 might be replicated as postdose value of Periods 1, 2, 3 and baseline value of Period 2, 3, 4. When serving as baseline of Periods 2, 3, 4, the recheck or unscheduled values after Day 11 of Periods 1, 2, 3 and prior to dosing of Periods 2, 3, 4 could be used as baseline.

## 7.5 Vital Signs (Blood Pressure, Pulse Rate, Respiration Rate, and Temperature)

Vital signs will be performed at the following time points:

**Table 7.5 Vital Signs Time Points** 

| | 1 | | 1 |
|-----------------|-------------------|------------|---------------|
| Period | Period Day | Study Hour | Assessment* |
| Screen | | | HR, BP, RR, T |
| 1 | Day -1 (check-in) | | HR, BP, RR, T |
| 1-4 | Day 1 | -0.75 | HR, BP, RR, T |
| 1-4 | Day 1 | 0.75, 2, 4 | HR, BP, RR |
| 1-4 | Day 2 | 24, 36 | HR, BP, RR |
| 1-4 | Day 3 | 48 | HR, BP, RR |
| 1-4 | Day 4 | 72 | HR, BP, RR |
| 1-4 | Day 5 | 96 | HR, BP, RR |
| 1-4 | Day 6 | 120 | HR, BP, RR |
| 1-4 | Day 11 | 240 | HR, BP, RR, T |
| End of | | | HR, BP, RR, T |
| Treatment/Early | | | |
| Termination | | | |

<sup>\*</sup> HR = Heart Rate, BP = Blood Pressure, RR = Respiration Rate,

Descriptive statistics will be reported for vital sign measurements (blood pressure, pulse, and respiration rate) and change from baseline by treatment and time point. Baseline is Day 1 predose and is the last non-missing predose measurement prior to dosing, including rechecks and unscheduled assessments. Postdose rechecks, unscheduled assessments, and ET results will not be used for calculation of descriptive statistics. All vital signs results will be listed by subject.

# 7.6 Safety ECG (Heart Rate, PR, QRS, QT, and QTcF [QT with Fridericia correction])

Single 12-lead ECGs will be performed at the following time points:

**Table 7.6: ECG Time Points** 

| Period | | Period Day | Study Hour |
|--------|-----|------------|-------------|
| Screen | | Screening | |
| | 1-4 | Day 1 | -0.75, 2, 4 |
| | 1-4 | Day 2 | 24, 36 |
| | 1-4 | Day 3 | 48 |

T = Temperature

Period Day 1 in Periods 2-4 is the same as Period Day 11 of the previous period.

| Period | Period Day | Study Hour |
|---|---|---|
| 1-4 | Day 4 | 72 |
| 1-4 | Day 5 | 96 |
| 1-4 | Day 6 | 120 |
| 1-4 | Day 11 | 240 |
| End of | · | |
| Treatment/Early | | |
| Termination | | |
| Period Day 1 in Periods 2-4 is the same as Period Day 11 of | | |

Period Day 1 in Periods 2-4 is the same as Period Day 11 of the previous period.

Descriptive statistics will be reported for ECG parameters and change from baseline by treatment and time point. Baseline is Day 1 predose and is the last non-missing predose measurement prior to dosing, including rechecks and unscheduled assessments. Postdose rechecks, unscheduled assessments, and ET results will not be used for calculation of descriptive statistics. All ECG interval parameters will be listed by subject and time point of collection with QTcF > 450 msec and change from baseline > 30 msec flagged.

#### 7.7 Concomitant Medications

All concomitant medications recorded during the study will be coded with the WHO Dictionary, Version 01-Mar-2019 b3 and listed.

## 7.8 Physical Examination

A full physical examination will be performed at screening. An abbreviated physical examination will be performed on Day 1 (prior to dosing of each period). Abnormal findings will be reported as medical history or adverse events by the clinical site. Physical examination results will be listed by subject and time point.

#### 8. SUMMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS

The analyses described in this SAP are aligned with those analyses described in the protocol.

## 9. SUMMARY TABLES AND FIGURES

Summary tables and figures are numbered following the International Council for Harmonization (ICH) structure but may be renumbered as appropriate during the compilation of the tables and figures for the CSR. Note that all summary tables and figures will be generated using SAS® Version 9.3 or higher.

## 9.1 In-text Summary Tables and Figures

The following is a list of table and figure titles that will be included in the text of the CSR. Tables and figures will be numbered appropriately during compilation of the CSR.

#### Section 10:

Table 10-1 Summary of Disposition (Safety Population)

## Section 11:

- Table 11-1 Demographic Summary (Safety Population)
- Table 11-2 Summary of Plasma LOXO-292 Pharmacokinetic Parameters
  Following Administration of a Single Oral Dose of CC mg
  LOXO-292 (Treatment A) and Single Oral Dose of mg LOXO292 (Treatment B) (Pharmacokinetic Population)
- Table 11-3 Summary of Plasma Moxifloxacin Pharmacokinetic Parameters Following Administration of a Single Oral Dose of Moxifloxacin (Treatment C) (Pharmacokinetic Population)
- Figure 11-1 Arithmetic Mean Plasma LOXO-292 Concentration-Time Profiles Following Administration of a Single Oral Dose of LOXO-292 (Treatment A) and Single Oral Dose of mg LOXO-292 (Treatment B) (Pharmacokinetic Population)
- Figure 11-2 Arithmetic Mean Plasma Moxifloxacin Concentration-Time Profile Following Administration of a Single Oral Dose of Moxifloxacin (Treatment C) (Pharmacokinetic Population)

#### Section 12:

Table 12-1 Treatment-Emergent Adverse Event Frequency by Treatment – Number of Subjects Reporting the Event (% of Subjects Dosed) (Safety Population)

#### 9.2 Section 14 Summary Tables and Figures

The following is a list of table and figure titles that will be included in Section 14 of the report. Table and figure titles may be renumbered as appropriate during the compilation of the report.

## 14.1 Demographic Data Summary Tables

#### 14.1.1 Demographic Tables

- Table 14.1.1.1 Summary of Disposition (Safety Population)
- Table 14.1.1.2 Disposition of Subjects (Safety Population)
- Table 14.1.1.3 Demographic Summary (Safety Population)

## 14.2 Pharmacokinetic Data Summary Tables and Figures

#### 14.2.1 LOXO-292

#### 14.2.1.1 Plasma LOXO-292 Tables

- Table 14.2.1.1.1 Plasma LOXO-292 Concentrations (ng/mL) Following Administration of a Single Oral Dose of Ing LOXO-292 (Treatment A) (Pharmacokinetic Population)
- Table 14.2.1.1.2 Plasma LOXO-292 Concentrations (ng/mL) Following Administration of a Single Oral Dose of mg LOXO-292 (Treatment B) (Pharmacokinetic Population)
- Table 14.2.1.1.3 Plasma LOXO-292 Concentrations (ng/mL) Following Oral Administration of LOXO-292 Matching Placebo (Treatment D) (Pharmacokinetic Population)
- Table 14.2.1.1.4 Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Oral Dose of LOXO-292 (Treatment A) (Pharmacokinetic Population)
- Table 14.2.1.1.5 Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Oral Dose of LOXO-292 (Treatment B) (Pharmacokinetic Population)
- Table 14.2.1.1.6 Intervals (Hours) Used for Determination of Plasma
  LOXO-292 Kel Values Following Administration of a
  Single Oral Dose of mg LOXO-292 (Treatment A) and
  Single Oral Dose of mg LOXO-292 (Treatment B)
  (Pharmacokinetic Population)

## 14.2.1.2 Plasma LOXO-292 Figures

- Figure 14.2.1.2.1 Mean (SD) Plasma LOXO-292 Concentration-Time
  Profiles Following Administration of a Single Oral Dose of
  mg LOXO-292 (Treatment A) and Single Oral Dose of
  mg LOXO-292 (Treatment B) (Linear Scale)
  (Pharmacokinetic Population)
- Figure 14.2.1.2.2 Mean Plasma LOXO-292 Concentration-Time Profiles
  Following Administration of a Single Oral Dose of
  LOXO-292 (Treatment A) and Single Oral Dose of mg
  LOXO-292 (Treatment B) (Linear Scale) (Pharmacokinetic
  Population)
- Figure 14.2.1.2.3 Mean Plasma LOXO-292 Concentration-Time Profiles Following Administration of a Single Oral Dose of mg

LOXO-292 (Treatment A) and Single Oral Dose of Communication (Semi-Log Scale) (Pharmacokinetic Population)

#### 14.2.2 Moxifloxacin

#### 14.2.2.1 Plasma Moxifloxacin Tables

- Table 14.2.2.1.1 Plasma Moxifloxacin Concentrations (ng/mL) Following Administration of a Single Oral Dose of Moxifloxacin (Treatment C) (Pharmacokinetic Population)
- Table 14.2.2.1.2 Plasma Moxifloxacin Pharmacokinetic Parameters
  Following Administration of a Single Oral Dose of mg
  Moxifloxacin (Treatment C) (Pharmacokinetic Population)
- Table 14.2.2.1.3 Intervals (Hours) Used for Determination of Plasma Moxifloxacin Kel Values Following Administration of a Single Oral Dose of mg Moxifloxacin (Treatment C) (Pharmacokinetic Population)

## 14.2.2.2 Plasma Moxifloxacin Figures

- Figure 14.2.2.2.1 Mean (SD) Plasma Moxifloxacin Concentration-Time
  Profile Following Administration of a Single Oral Dose of
  Comp Moxifloxacin (Treatment C) (Linear Scale)
  (Pharmacokinetic Population)
- Figure 14.2.2.2.2 Mean Plasma Moxifloxacin Concentration-Time Profile
  Following Administration of a Single Oral Dose of
  Moxifloxacin (Treatment C) (Linear Scale)
  (Pharmacokinetic Population)
- Figure 14.2.2.2.3 Mean Plasma Moxifloxacin Concentration-Time Profile
  Following Administration of a Single Oral Dose of Moxifloxacin (Treatment C) (Semi-Log Scale)
  (Pharmacokinetic Population)

## 14.3 Safety Data Summary Tables

#### 14.3.1 Displays of Adverse Events

- Table 14.3.1.1 Treatment-Emergent Adverse Event Frequency by Treatment
   Number of Subjects Reporting Events (% of Subject
  Dosed) (Safety Population)
- Table 14.3.1.2 Treatment-Emergent Adverse Event Frequency by
  Treatment, Severity Grade, and Relationship to Study Drugs
   Number of Subjects Reporting Events (Safety Population)

## 14.3.2 Listings of Deaths, other Serious and Significant Adverse Events

Table 14.3.2.1 Serious Adverse Events (Safety Population)

<If no serious adverse event occurred, a statement 'There was no serious adverse event recorded during the study.' will be added.>

## 14.3.3. Narratives of Deaths, other Serious and Certain other Significant Adverse Events

## 14.3.4. Abnormal Laboratory Value Listing (each patient)

- Table 14.3.4.1 Out-of-Range Values and Recheck Results Serum Chemistry (Safety Population)
- Table 14.3.4.2 Out-of-Range Values and Recheck Results Hematology and Coagulation
- Table 14.3.4.3 Out-of-Range Values and Recheck Results Urinalysis
- Table 14.3.4.4 Clinically Significant Laboratory and Corresponding Results (Safety Population)

# 14.3.5. Displays of Other Laboratory, Vital Signs, Electrocardiogram, Physical Examination, and Other Safety Data

- Table 14.3.5.1 Clinical Laboratory Summary and Change From Baseline Serum Chemistry (Safety Population)
- Table 14.3.5.2 Clinical Laboratory Shift From Baseline Serum Chemistry (Safety Population)
- Table 14.3.5.3 Clinical Laboratory Summary and Change From Baseline Hematology and Coagulation (Safety Population)
- Table 14.3.5.4 Clinical Laboratory Shift From Baseline Hematology and Coagulation (Safety Population)
- Table 14.3.5.5 Clinical Laboratory Summary and Change From Baseline Urinalysis (Safety Population)
- Table 14.3.5.6 Clinical Laboratory Shift From Baseline Urinalysis (Safety Population)
- Table 14.3.5.7 Vital Sign Summary and Change From Baseline (Safety Population)
- Table 14.3.5.8 12-Lead Electrocardiogram Summary and Change From Baseline (Safety Population)

## 9.3 Section 16 Data Listings

Note: Virology test results (Hepatitis and HIV) that are provided by the clinical laboratory will not be presented in subject data listings and will not be included in the database transfer.

Data listings are numbered following the ICH structure but may be renumbered as appropriate during the compilation of the tables and figures for the CSR. The following is a list of appendix numbers and titles that will be included as data listings:

## **16.1** Study Information

Appendix 16.1.9 Statistical Methods

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

## 16.2. Subject Data Listings

## **16.2.1.** Subject Discontinuation

Appendix 16.2.1 Subject Discontinuation (Safety Population)

#### **16.2.2.** Protocol Deviations

Appendix 16.2.2 Protocol Deviations

Note: Protocol deviations will be provided by the clinical study manager as Microsoft Excel file and read into the SDTM to generate the data listing.

## 16.2.3. Subjects Excluded from Pharmacokinetic Analysis

Appendix 16.2.3 Subjects Excluded from Pharmacokinetic Analysis

Note: Appendix 16.2.3 is generated in MS Word for inclusion in the CSR.

## 16.2.4 Demographic Data

| Appendix 16.2.4.1 | Demographics (Safety Population) |
|-------------------|--------------------------------------------------|
| Appendix 16.2.4.2 | Updated Informed Consent (Safety Population) |
| Appendix 16.2.4.3 | Physical Examination (Safety Population) |
| Appendix 16.2.4.4 | Medical and Surgical History (Safety Population) |
| Appendix 16.2.4.5 | Nicotine Use (Safety Population) |

## 16.2.5. Compliance and Drug Concentration Data

| Appendix 16.2.5.1.1 | Inclusion Criteria |
|---------------------|-----------------------------------------|
| Appendix 16.2.5.1.2 | Exclusion Criteria |
| Appendix 16.2.5.2 | Subject Eligibility (Safety Population) |
| Appendix 16.2.5.3.1 | Check-in Criteria |
| Appendix 16.2.5.3.2 | Check-in Responses (Safety Population) |
| Appendix 16.2.5.4.1 | Test Compound Description |

| Appendix 16.2.5.4.2 | Test Compound Administration Times (Safety Population) |
|---|---|
| Appendix 16.2.5.5 | PK Blood Draw Times (Safety Population) |
| Appendix 16.2.5.6 | Meal Times (Safety Population) |
| Appendix 16.2.5.7 | Prior and Concomitant Medications (Safety Population) |
| 16.2.6 Individual | Pharmacokinetic Response Data |
| Appendix 16.2.6.1 | Individual Plasma LOXO-292 Concentration Versus Time Profiles Following Administration of a Single Oral Dose of CO mg LOXO-292 (Treatment A) and Single Oral Dose of CO mg LOXO-292 (Treatment B) for Subject X (Linear and Semi-Log Scales) |
| Appendix 16.2.6.2 | Individual Plasma Moxifloxacin Concentration Versus Time Profiles Following Administration of a Single Oral Dose of [CC] mg Moxifloxacin (Treatment C) for Subject X (Linear and Semi-Log Scale) |
| 16.2.7 Adverse Ev | rents Listings |
| Appendix 16.2.7.1 | Adverse Events (I of II) (Safety Population) |
| Appendix 16.2.7.2 | Adverse Events (II of II) (Safety Population) |
| Appendix 16.2.7.3 | Adverse Event Non-Drug Therapy (Safety Population) |
| Appendix 16.2.7.4 | Adverse Event Preferred Term Classification (Safety Population) |
| 16.2.8 Listings of Safety Obse | Individual Laboratory Measurements and Other ervations |
| Appendix 16.2.8.1.1 | Clinical Laboratory Report - Serum Chemistry (Safety Population) |
| Appendix 16.2.8.1.2 | Clinical Laboratory Report - Hematology and<br>Coagulation (Safety Population) |
| Appendix 16.2.8.1.3 | Clinical Laboratory Report - Urinalysis (Safety Population) |
| Appendix 16.2.8.1.4 | Clinical Laboratory Report - Urine Drug Screening (Safety Population) |
| Appendix 16.2.8.1.5 | Clinical Laboratory Report - Comments (Safety Population) |
| Appendix 16.2.8.2 | Vital Signs (Safety Population) |
| Appendix 16.2.8.3 | 12-Lead Electrocardiogram (Safety Population) |
| Appendix 16 2 8 4 | Holter Monitoring Times (Safety Population) |

Appendix 16.2.8.5 Phone Call (Safety Population)

## 10. TABLE AND FIGURE SHELLS

The following table shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the tables and figures that will be presented and included in the final CSR. Unless otherwise noted, all in-text tables will be presented in Times New Roman font size 8 and post-text tables in Courier New size font 9. These tables will be generated according to the ADaM Model 2.1 and ADaM implementation guide 1.1.

Actual treatment sequence will be used unless the column header uses the reference randomized sequence. Period Day will be used unless there is a footnote describing that the day referenced is using Period 1 Day 1 (ie, AE listing).

#### 10.1 **In-text Table Shells**

**Summary of Disposition (Safety Population) Table 10-1** 

| Disposition | Randomized Sequence | | | | Overall |
|---|---|---|---|---|---|
| | ABCD | BCDA | CDAB | DABC | Overall |
| Enrolled | XX (100%) | XX (100%) | XX (100%) | XX (100%) | XX (100%) |
| Completed Study | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Discontinued Early | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| <reason1></reason1> | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| <reason2></reason2> | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |

Treatment A: <>
Treatment B: <>

Treatment C: <>

Treatment D: <>

Source: Table 14.1.1.1

Program: /CAXXXXX/sas\_prg/stsas/intext/t\_disp.sas DDMMMYYYY HH:MM

**Table 11-1 Demographic Summary (Safety Population)** 

| | | Randomized Sequence | | | | |
|---|---|---|---|---|---|---|
| Trait | | ABCD | BCDA | CDAB | DABC | Study Overall |
| Sex | Male | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Female | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Race | Asian | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Black or African<br>American | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | White | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Ethnicity | Hispanic or Latino | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Not Hispanic or Latino | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Age* (yr) | n | XX | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | Minimum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Maximum | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Height (cm) | n | XX | XX | XX | XX | XX |
| | Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X.XX |
| | Minimum | XXX | XXX | XXX | XXX | XXX |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | Maximum | XXX | XXX | XXX | XXX | XXX |

<sup>\*</sup> Age is calculated from the date of first dosing.

BMI = Body mass index

Source: Table 14.1.1.3

Program: /CAXXXXX/sas\_prg/stsas/intexttest/t\_dem.sas DDMMMYYYY HH:MM

**Programmer Note:** Weight (kg) and BMI (kg/m²) will also be summarized in the table above.

In-text Tables 11-2 and 11-3 will be in the following format:

Table 11-2 Summary of Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Oral Dose of Total mg LOXO-292 (Treatment A) and Single Oral Dose of Total mg LOXO-292 (Treatment B) (Pharmacokinetic Population)

| Pharmacokinetic Parameters | mg LOXO-292 | mg LOXO-292 |
|---|---|---|
| Param1 (units) | XXX.X (XX.X) [n=xx] $XXX.X (XX.X) [n=xx]$ | |
| Param2 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param3 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| Param4 (units) | XXX.X (XX.X) [n=xx] | XXX.X (XX.X) [n=xx] |
| mg LOXO-292: mg LOXO-292 mg LOXO-292 mg LOXO-292 mg LOXO-292 matching placebo local mg mg matching placebo local mg LOXO-292: mg LOXO-292: mg LOXO-292 | | |
| AUC and Cmax values are presented as geometric mean (geometric CV%). | | |
| Tmax values are presented as median (min, max). | | |
| Other parameters are presented as arithmetic mean (± SD). | | |
| Source: Tables 14.2.1.1.4 and 14.2.1.1.5 | | |

## **Notes for Generating the Actual Table:**

## Presentation of Data:

- The following PK parameters will be presented in the following order: AUC0-t, AUC0-inf, AUC%extrap, Cmax, Tmax, Kel, and t½;
- Table 11-2 source: Tables 14.2.1.1.4 and 14.2.1.1.5
- Table 11-3 source: Table 14.2.2.1.2
- n will be presented as an integer (with no decimal);
- Summary statistics will be presented with same precision as defined in post-text shells

Program: /CAXXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMYYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam\_intext\_pkparam.sas DDMMYYYYY HH:MM

Table 12-1 Treatment-Emergent Adverse Event Frequency by Treatment – Number of Subjects Reporting the Event (% of Subjects Dosed) (Safety Population)

| | Treatment | | | | Overall |
|---|---|---|---|---|---|
| Adverse Events* | A | В | C | D | |
| Number of Subjects Dosed | XX (100%) | XX (100%) | XX (100%) | Similar to Previous<br>Column | XX (100%) |
| Number of Subjects With TEAEs | XX (XX%) | XX (XX%) | XX (XX%) | | XX (XX%) |
| Number of Subjects Without TEAEs | XX (XX%) | XX (XX%) | XX (XX%) | | XX (XX%) |
| System Organ Class 1 | X ( X%) | X ( X%) | X ( X%) | | X ( X%) |
| Preferred Term 1 | X ( X%) | X ( X%) | X ( X%) | | X ( X%) |
| Preferred Term 2 | X ( X%) | X ( X%) | X ( X%) | | X ( X%) |
| System Organ Class 2 | X ( X%) | X ( X%) | X ( X%) | | X ( X%) |
| Preferred Term 1 | X ( X%) | X ( X%) | X ( X%) | | X ( X%) |
| Preferred Term 2 | X ( X%) | X ( X%) | X ( X%) | | X ( X%) |

<sup>\*</sup> Adverse events are coded using MedDRA® Version 22.0 by System Organ Class and Preferred Term.

Although a subject may have had 2 or more clinical adverse experiences, the subject is counted only once within a category. The same subject may appear in different categories.

If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity under the same treatment group.

Treatment A: <>
Treatment B: <>
Treatment C: <>
Treatment D: <>

Source: Table 14.3.1.1

Program: /CAXXXXX/sas\_prg/stsas/intexttest/t\_ae.sas DDMMMYYYY HH:MM

Programmer Note: Sort by decreasing frequency of system organ class and by preferred term within a system organ class of Overall column.

TEAE = Treatment-emergent Adverse event

## 10.2 Figures Shells

In-text Figures 11-1 and 11-2 and Figures 14.2.1.2.2 and 14.2.2.2.2 will be in the following format:

Figure 11-1 Arithmetic Mean Plasma LOXO-292 Concentration-Time Profiles Following Administration of a Single Oral Dose of mg LOXO 292 (Treatment A) and Single Oral Dose of mg LOXO-292 (Treatment B) (Pharmacokinetic Population)



Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

Statistical Analysis Plan, 28 June 2019

## **Notes for Generating the Actual Mean Figure:**

- Figures 11-1 and 14.2.1.2.2:
  - o Legend will be:

    - Treatment A: CC mg LOXO-292
       Treatment B: CC mg LOXO-292
  - o Y-axis label will be "Plasma LOXO-292 Concentration (ng/mL)"
  - X-axis label will be "Hours Postdose (hr) from LOXO-292 Dose"
  - o Add in footnote: LLOQ value for LOXO-292 is 1.00 ng/mL
- Figures 11-2 and 14.2.2.2.2:
  - o Legend will be:
    - CCI mg moxifloxacin
  - o Y-axis label will be "Plasma Moxifloxacin Concentration (ng/mL)"
  - X-axis label will be "Hours Postdose (hr) from Moxifloxacin Dose"
  - Add in footnote: LLOQ value for moxifloxacin is 25 ng/mL.

Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMYYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYYY HH:MM

Figures 14.2.1.2.1 and 14.2.2.2.1 will be in the following format:

Figure 14.2.1.2.1 Arithmetic Mean (SD) Plasma LOXO-292 Concentration-Time Profiles Following Administration of a Single Oral Dose of mg LOXO 292 (Treatment A) and Single Oral Dose of mg LOXO-292 (Treatment B) (Pharmacokinetic Population)



Treatments B and C are shifted to the right for ease of reading

Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

## Notes for Generating the Actual Mean Figure:

- Figures 14.2.1.2.1:
  - o Legend will be:

    - Treatment A: CC mg LOXO-292
       Treatment B: CC mg LOXO-292
  - o Y-axis label will be "Plasma LOXO-292 Concentration (ng/mL)"
  - X-axis label will be "Hours Postdose (hr) from LOXO-292 Dose"
  - o Add in footnote: LLOQ value for LOXO-292 is 1.00 ng/mL
- Figures 14.2.2.2.1:
  - o Legend will be:
    - ccl mg moxifloxacin
  - o Y-axis label will be "Plasma Moxifloxacin Concentration (ng/mL)"
  - X-axis label will be "Hours Postdose (hr) from Moxifloxacin Dose"
  - Add in footnote: LLOQ value for moxifloxacin is 25 ng/mL.

Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMYYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYYY HH:MM
Figures 14.2.1.2.3 and 14.2.2.2.3 will be in the following format:

Figure 14.2.1.2.3 Mean Plasma LOXO-292 Concentration-Time Profiles Following Administration of a Single Oral Dose of mg LOXO-292 (Treatment A) and Single Oral Dose of mg LOXO-292 (Treatment B) (Semi-Log Scale) (Pharmacokinetic Population)



Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

## **Notes for Generating the Actual Mean Figure:**

- Figures 14.2.1.2.3:
  - o Legend will be:

    - Treatment A: CC mg LOXO-292
       Treatment B: CC mg LOXO-292
  - o Y-axis label will be "Plasma LOXO-292 Concentration (ng/mL)"
  - X-axis label will be "Hours Postdose (hr) from LOXO-292 Dose"
  - o Add in footnote: LLOQ value for LOXO-292 is 1.00 ng/mL
- Figures 14.2.2.2.3:
  - o Legend will be:
    - moxifloxacin
  - o Y-axis label will be "Plasma Moxifloxacin Concentration (ng/mL)"
  - X-axis label will be "Hours Postdose (hr) from Moxifloxacin Dose"
  - Add in footnote: LLOQ value for moxifloxacin is 25 ng/mL.

Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMYYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYYYY HH:MM Appendix 16.2.6.1 and 16.2.6.2 will be in the following format:

## Appendix 16.2.6.1

Individual Plasma LOXO-292 Concentration Versus Time Profiles Following Administration of a Single Oral Dose of mg LOXO-292 (Treatment A) and Single Oral Dose of LOXO-292 (Treatment B) for Subject X (Linear and Semi-Log Scales)



Program: /CAXXXXX/sas\_prg/pksas/adam\_indgraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/indgraph-all.sas DDMMMYYY HH:MM

## Notes for Generating the Actual Individual Figure:

- Appendix 16.2.6.1:
  - Legend will be:

    - Treatment A: CCl mg LOXO-292 Treatment B: CCl mg LOXO-292
  - o Y-axis label will be "Plasma LOXO-292 Concentration (ng/mL)"
  - o X-axis label will be "Hours Postdose (hr) from LOXO-292 Dose"
  - o Add in footnote: LLOQ value for LOXO-292 is 1.00 ng/mL
- Appendix 16.2.6.2:
  - o Legend will be:
    - mg moxifloxacin
  - o Y-axis label will be "Plasma Moxifloxacin Concentration (ng/mL)"
  - o X-axis label will be "Hours Postdose (hr) from Moxifloxacin Dose"
  - o Add in footnote: LLOQ value for moxifloxacin is 25 ng/mL.

Program: /CAXXXXX/sas\_prg/pksas/indgraph-all.sas DDMMMYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam\_indgraph.sas DDMMMYYYY HH:MM

## 10.3 Post-text Table Shells

Table 14.1.1.1 Summary of Disposition (Safety Population)

Page X of X

| Randomized | Sequence |
|------------|----------|

| Disposition | ABCD | BCDA | CDAB | DABC | Overall |
|--------------------|------|------|------|------|---------|
| Enrolled | XX | XX | XX | XX | XX |
| Completed | XX | XX | XX | XX | XX |
| Discontinued Early | XX | XX | XX | XX | XX |
| Reason 1 | XX | XX | XX | XX | XX |
| Reason 2 | XX | XX | XX | XX | XX |
| Reason 3 | XX | XX | XX | XX | XX |
| etc. | | | | | |

Note: Treatment A: < >

Treatment B: < >

Treatment C: < >

Treatment D: < >

Page X of X

Table 14.1.1.2 Disposition of Subjects (Safety Population)

| Cubicat | Dandominod | | Dosed | l Period | l | Study Completion | |
|---|---|---|---|---|---|---|---|
| | Randomized<br>Sequence | 1 | 2 | 3 | 4 | Status | Date |
| XXX-XXX<br>XXX-XXX | | Yes<br>Yes | Yes<br>Yes | Yes<br>Yes | Yes<br>No | Completed Study<br>Terminated Study Prematurely | DDMMYYYY<br>DDMMYYYY |

Note: Treatment A: < >

Treatment B: < >

Treatment C: < >

Treatment D: < >


Table 14.1.1.3 Demographic Summary (Safety Population)

| | | Ran | domized | | | |
|---|---|---|---|---|---|---|
| Trait | | ABCD | BCDA | CDAB | DABC | Study<br>Overall |
| Sex | Male<br>Female | X ( XX%)<br>X ( XX%) | | to col | umn ABCD | for all other columns> |
| Race | Asian<br>Black or African American<br>White | X ( XX%)<br>X ( XX%)<br>X ( XX%) | | | | |
| Ethnicity | Hispanic or Latino<br>Not Hispanic or Latino | | | | | |
| Age* (yr) | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.X<br>X.XX<br>XX<br>XX.X | | | | |
| Height (cm) | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.X<br>XX.XX<br>XX<br>XX.X | | | | |

**Programmer Note:** Also include weight (kg) and BMI (kg/m²)

Note: \* Age is calculated from the date of first dosing.  ${\tt BMI} = {\tt Body} \ {\tt mass} \ {\tt index}$ 

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMYYYYY HH:MM

## Tables 14.2.1.1.1, 14.2.1.1.2, 14.2.1.1.3, and 14.2.2.1.1 will be in the following format:

Table 14.2.1.1.1 Plasma LOXO-292 Concentrations (ng/mL) Following Administration of a Single Oral Dose of [CC] mg LOXO-292 (Treatment A) (Pharmacokinetic Population)

| Subject | Treatment | Chd. | | | | Samp | ole Times | (hr) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Treatment | Study | | | | | | | | | _ |
| Number | Sequence | Period | Predose | XX | XX | XX | XX | XX | XX | XX | XX |
| XXX-XXX | XXXX | Х | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| XXX-XXX | XXXX | X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| XXX-XXX | XXXX | X | BLQ | XX | XX | XX | XX | XX | XX | XX | XX |
| n | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mean | | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | | | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SEM | | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Median | | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Maximum | | | XX | XX | XX | XX | XX | XX | XX | XX | XX |

For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of 1 ng/mL are treated as 0 before the first quantifiable concentration and as missing elsewhere.

<sup>. =</sup> Value missing or not reportable.

## **Notes for Generating the Actual Table:**

#### Presentation of Data:

- Present the subject number in the following format: XXX-XXX
- Concentrations will be presented to same precision as in the bioanalytical data.
- Summary statistics presentation with respect to the precision of the bioanalytical data: n = integer; Mean and Median +1; SD and SEM +2, Min and Max +0, CV% to 1 decimal

## Programmer Note:

- PK Time points are:
  - o LOXO-292 Tables 14.2.1.1.1, 14.2.1.1.2, and 14.2.1.1.3: predose and 0.25, 0.5, 0.75, 1.5, 2, 2.5, 3, 4, 7, 9, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, and 240 hours postdose.
  - o Moxifloxacin Table 14.2.2.1.1: predose and 0.25, 0.5, 0.75, 1.5, 2, 2.5, 3, 4, 7, 9, 12, and 24 hours postdose.

Program: /CAXXXX/sas\_prg/pksas/pk-conc-tables.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/pk-conc-tables-sig.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/adam\_conc.sas DDMMYYYY HH:MM

# Tables 14.2.1.1.4, 14.2.1.1.5 and 14.2.2.1.2 will be in the following format:

Table 14.2.1.1.4 Plasma LOXO-292 Pharmacokinetic Parameters Following Administration of a Single Oral Dose of CT mg LOXO-292 (Treatment A) (Pharmacokinetic Population)

| | | eters | Param | | | | | |
|---|---|---|---|---|---|---|---|---|
| parame | param5 | param4 | param3 | param2 | param1 | Study | Treatment | Subject |
| (units) | (units) | (units) | (units) | (units) | (units) | Period | Sequence | Number |
| X.XXX | XX.X | XXX | XXX | X.XX | XXX | X | XXXX | XXX-XXX |
| X.XXX | XX.X | XXX | XXX | X.XX | XX.X | X | XXXX | XXX-XXX |
| X.XXX | XX.X | XXX | XXX | X.XX | XXX | X | XXXX | XXX-XXX |
| X.XXX | XX.X | XXX | XXX | X.XX | XX.X | X | XXXX | XXX-XXX |
| X.XXX | XX.X | XXX | XXX | X.XX | XX.X | X | XXXX | XXX-XXX |
| X.XXX | XX.X | XXX | XXX | X.XX | X.XX | X | XXXX | XXX-XXX |
| X.XXX | XX.X | XXX | XXX | X.XX | XXX | X | XXXX | XXX-XXX |
| XX | XX | XX | XX | XX | XX | | | n |
| X.XXXX | XX.XX | XXX.X | XXX.X | X.XXX | XXX.X | | | Mean |
| XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | | | SD |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | | | CV% |
| XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | | | SEM |
| X.XXX | XX.X | XXX | XXX | X.XX | XX.X | | | Minimum |
| X.XXXX | XX.XX | XXX.X | XXX.X | X.XXX | XX.XX | | | Median |
| X.XXX | XX.X | XXX | XXX | X.XX | XXX | | | Maximum |
| X.XXXX | XX.XX | XXX.X | XXX.X | X.XXX | XXX.X | | | Geom Mean |
| XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | | | Geom CV% |

<sup>. =</sup> Value missing or not reportable.

## **Notes for Generating the Actual Table:**

#### Presentation of Data:

- Present the subject number in the following format: XXX-XXX;
- The following PK parameters will be presented in the following order: AUC0-t, AUC0-inf, AUC%extrap, Cmax, Tmax, Kel, and t½;
- n will be presented as an integer (with no decimal);
- Parameter values for exposure-based parameters (i.e. AUCs, AUC%extrap, and Cmax) will be presented with 3 significant figures.
  - O Summary statistics for exposure parameters will be presented as: Mean, Median, and Geom Mean +1; SD and SEM +2, Min and Max +0 with respect to the number of significant figures.
- Values for time-based parameters (i.e. Tmax, and  $t\frac{1}{2}$ ) will be presented with 2 decimals.
  - Summary statistics for time-based parameters will be presented as: Mean, Median, and Geom Mean +1; SD and SEM +2, Min and Max +0 with respect to the number of decimals.
- Values for rate constants (i.e. Kel) will be presented with 3 significant figures.
  - O Summary statistics for Kel will be presented as: Mean, Median, and Geom Mean +1; SD and SEM +2, Min and Max +0 with respect to the number of significant figures.
- CV% and Geom CV% for all parameters will be presented with 1 decimal
- Table 14.2.1.1.4, 14.2.1.1.5 will be for LOXO-292 and Table 14.2.2.1.2 will be for moxifloxacin

Program: /CAXXXX/sas\_prg/pksas/pk-tables.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/adam\_pkparam.sas DDMMYYYY HH:MM

## Tables 14.2.1.1.6 and 14.2.2.1.3 will be in the following format:

Table 14.2.1.1.6 Intervals (Hours) Used for Determination of Plasma LOXO-292 Kel Values Following Administration of a Single Oral Dose of [60] mg LOXO-292 (Treatment A) and Single Oral Dose of [60] mg LOXO-292 (Treatment B) (Pharmacokinetic Population)

| Subject | Treatment | Treatm | ent A | ] | Treatment B | | |
|---|---|---|---|---|---|---|---|
| Number | Sequence | Interval | R2 | n | Interval | R2 | n |
| XXX-XXX | XXXX | XX.X - XX.X | x.xxx | X | xx.x - xx.x | x.xxx | X |
| XXX-XXX | XXXX | xx.x - xx.x | X.XXX | X | XX.X - XX.X | X.XXX | X |
| XXX-XXX | XXXX | XX.X - XX.X | X.XXX | X | XX.X - XX.X | X.XXX | X |

Treatment A: CCI mg LOXO-292 (CCICCI mg CCI mg LOXO-292 matching placebo (CCI mg mg matching placebo CCI administered at Hour 0 on Day 1

Treatment B: CC mg LOXO-292 (CC) CC mg CC mg CC mg administered at Hour 0 on Day 1

R2 = Coefficient of determination

n = Number of points used in Kel calculation

. = Kel value not reportable.

## **Notes for Generating the Actual Table:**

#### Presentation of Data:

- Present the subject number in the following format: XXX-XXX
- Interval start and stop times will be presented to 1 decimal or 3 significant figures minimum;
- R2 will be presented to 3 decimals;
- n will be presented as an integer (with no decimal)

Program: /CAXXXXX/sas\_prg/pksas/kel-tables-xover.sas DDMMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam\_kel.sas DDMMMYYYY HH:MM


Table 14.3.1.1 Treatment-Emergent Adverse Event Frequency by Treatment - Number of Subjects Reporting Events (% of Subject Dosed) (Safety Population)

| | Treatment | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| TE Adverse Event* | | A | | В | С | | D | Overall |
| Number of Subjects Dosed | | (100%) | | (100%) | X(100%) | X(10 | 00%) | <similar td="" to<=""></similar> |
| Number of Subjects with TE Adverse Events<br>Number of Subjects without TE Adverse Events | X | (XX%)<br>(XX%) | X | (XX%) | X (XX%) | X (Σ<br>X (Σ | | previous columns> |
| Nervous system disorders | X | (XX%) | X | (XX%) | X (XX%) | Χ (Σ | <br>⟨X%) | |
| Dizziness | Χ | (XX%) | X | (XX%) | X (XX%) | Χ (Σ | (X%) | |
| Headache | Χ | (XX%) | X | (XX%) | X (XX%) | Χ (Σ | (X%) | |
| Presyncope | Χ | (XX%) | X | (XX%) | X (XX%) | Χ (Σ | (X%) | |
| Respiratory, thoracic and mediastinal disorders | Χ | (XX%) | X | (XX%) | X (XX%) | Χ (Σ | (X%) | |
| Dry throat | Χ | (XX%) | X | (XX%) | X (XX%) | Χ (Σ | ⟨X%) | |
| Oropharyngeal pain | Χ | (XX%) | X | (XX%) | X (XX%) | X (X | (X%) | |
| Sinus congestion | Χ | (XX%) | X | (XX%) | X (XX%) | Χ (Σ | ⟨X%) | |
| Sneezing | Χ | (XX%) | X | (XX%) | X (XX%) | Χ (Σ | ⟨X%) | |
| General disorders and administration site conditions | Χ | (XX%) | X | (XX%) | X (XX%) | Χ (Σ | ⟨X%) | |
| Fatigue | Χ | (XX%) | X | (XX%) | X (XX%) | Χ (Σ | (X%) | |
| Thirst | Χ | (XX%) | Х | (XX%) | X (XX%) | X (X | (X%) | |
| etc. | | | | | | | | |

Note: \* Adverse events are classified according to the MedDRA Version 22.0 by System Organ Class and Preferred Term.

If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity under the same treatment group.

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Statistical Analysis Plan, 28 June 2019


TE = Treatment-emergent

Programmer Note: Sort by decreasing frequency of system organ class and by preferred term within a system organ class of Overall column. For each subject, please sort the AEs with same verbatim and preferred term by onset date/time. For any pair (e.g., AE\_S1, AE\_S2) of these AEs (for same subject, same verbatim and preferred term), if the onset date/time of AE\_S2 = resolved date/time of AE\_S1 and the grade of AE\_S2 < the grade level of AE\_S1, then mark the AE\_S2 with a flag like EVAUL\_FLG ="N". Then, for AE analysis (summary tables), please exclude the ones with EVAUL\_FLG ="N". Won't repeat this comment again.


Table 14.3.1.2 Treatment-Emergent Adverse Event Frequency by Treatment, Severity Grade, and Relationship to Study Drugs - Number of Subjects Reporting Events (Safety Population)

| | Treat- | Number of<br>Subjects with<br>Adverse Events | | | - | y Grade | | | ip to LOXO-292 | Relationship to Moxifloxacin | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| TE Adverse Event* | | | 1 | 2 | 3 | 4 | 5 | Related | Not Related | Related | Not Related |
| Dizziness | A | X | X | X | Χ | X | X | X | X | X | X |
| Dry eye | В | X | X | X | X | X | X | X | X | X | X |
| Dry mouth | A | X | X | X | X | X | X | X | X | X | X |
| - | С | X | X | X | X | X | X | X | X | X | X |
| Dry throat | D | X | X | X | X | X | X | X | X | X | X |
| Ear pain | A | X | X | X | X | X | X | X | X | X | X |
| Fatigue | D | X | Χ | Χ | Χ | Χ | Χ | X | X | X | X |
| Treatment A | | XX | X | X | Χ | X | X | X | X | X | X |
| Treatment B | | XX | X | X | X | X | X | X | X | X | X |
| Treatment C | | XX | X | X | X | X | X | X | X | X | X |
| Treatment D | | XX | X | X | X | X | X | X | X | X | X |
| Overall | | XX | Χ | Χ | Χ | Χ | Χ | X | X | X | X |

Note: \* Adverse events are classified according to MedDRA Version 22.0 by System Organ Class and Preferred Term.

TE = Treatment-emergent; AE = Adverse event

Severity Grade: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately lifethreatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE

Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection. If a TEAE decreased in severity grade, the new TEAE record with less severity was counted as the same TEAE event of the previous record with worse severity under the same treatment group.

When a subject experienced the same TEAE at more than one level of severity during a treatment period, only the most severe one was counted.

When a subject experienced the same TEAE at more than one level of drug relationship during a treatment period, only the one related to study drugs was counted.

Treatment A: < >

Treatment B: < >

Treatment C: < >

Treatment D: < >

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Page X of X

#### Table 14.3.2.1 Serious Adverse Events (Safety Population)

| Subject | Treat- | | Adverse | PT*/ | On | set/Resolut | ion | | Severity | | | | | Relationship to LOXO-292/ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | ment | TE?^ | Event | SOC | Day | Date | Time | Freq! | Grade | Act~ | Ser@ | Outcome | Moxifloxacin | Moxifloxacin |
| XXX-XXX | X | Yes | XXXXXXX | XXXXXXX/<br>XXXXXXXX | XX/<br>XX | DDMMYYYY/<br>DDMMYYYYY | | Inter. | X | Х | NS | Resolved | XXXXXXXXX/<br>XXXXXXXXX | XXXXXXXXX/<br>XXXXXXXXX |

TE^ = Treatment-emergent; PT = Preferred Term; SOC = System Organ Class, Onset day is relative to Period 1 Day 1.

Freq! represents Frequency: SI = Single Episode, Inter. = Intermittent, Cont. = Continuous

Act~: 1 = None, 2 = Medication Required, 3 = Non-drug therapy required, 4 = Medication and Non-drug therapy required, 5 = Subject Withdrawn, 6 = Hospitalization, 7 = Other

Ser@ represents Serious: NS = Not Serious

Severity/Intensity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately life-threatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE

Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection. Treatment A: < >

Note: \* Adverse events are classified according to MedDRA Version 22.0 by System Organ Class and Preferred Term.

Treatment B: < >
Treatment C: < >

Treatment D: < >

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYYY HH:MM

Programmer Note: if there are no serious adverse events reported, there will be just one table (Table 14.3.2.1) with the statement "There was no serious adverse event recorded during the study."

Statistical Analysis Plan, 28 June 2019


## Tables 14.3.4.2-14.3.4.3 will have the following format.


Table 14.3.4.1 Out-of-Range Values and Recheck Results - Serum Chemistry (Safety Population)

| Subject<br>Number | Age\$/<br>Sex | Study<br>Period | Day | Date | Parameter1<br>< Range><br>(Unit) | Parameter2<br>< Range><br>(Unit) | Parameter3<br>< Range><br>(Unit) | Parameter4<br>< Range><br>(Unit) | Parameter5<br>< Range><br>(Unit) |
|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XX/M | Screen | | DDMMYYYY | XX HN | | | | XX HN |
| | | 1 | -X | DDMMYYYY | | XX LN | XX HYR- | | |
| | | 2 | X | DDMMYYYYY | | | | XX HN^+ | |
| | | | X | DDMMYYYYY | XX LY- | | | | |
| | | | X | DDMMYYYYY | | XX LY- | | | |

Programmer Note: Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for. Arrange alphabetically by lab test name.

Note: \$ Age is calculated from the date of first dosing

Abnormal flag: H = Above Reference Range, L = Below Reference Range

Computer Clinical significance: N = Not Clinically Significant, Y = Clinically Significant

PI Interpretation: - = Not Clinically Significant, + = Clinically Signficant, R = To be Rechecked, ^ = Will be Retested at a Later Event

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM


Table 14.3.4.4 Clinically Significant Laboratory and Corresponding Results (Safety Population)

| Subject<br>Number | | | Day | Date | Time | Department | Test | Result | Reference Range | Unit |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XX/X | Х | X | DDMMYYYY | HH:MM:SS | Serum Chemistry | Cholesterol | XXX | X - X | mg/dL |
| | | | X | DDMMYYYYY | HH:MM:SS | Serum Chemistry | Cholesterol | XXX HYR+ | X - X | mg/dL |
| | | | X | DDMMYYYY | HH:MM:SS | Serum Chemistry | Cholesterol | XXX HY- | X - X | mg/dL |
| | | | X | DDMMYYYYY | HH:MM:SS | Serum Chemistry | Cholesterol | XXX HN | X - X | mg/dL |

Programmer Note: All time points for a subject/test with at least one value deemed as CS by the PI will be presented in this table.

If there were no CS values as deemed by PI (i.e., no "CS" or "Clinically Significant" in the PI flag [3rd or 4th field] in the laboratory dataset), then this table will contain only the statement: "There were no laboratory values deemed clinically significant by the PI in the study."

Note: \$ Age is calculated from the date of first dosing
H = Above Reference Range, L = Below Reference Range

Computer: N = Not Clinically Significant, Y = Clinically Significant

PI Interpretation: - = Not Clinically Significant, R = To be Rechecked, ^ = Will be Retested at a Later Event, + = Clinically Significant

## Tables 14.3.5.1, 14.3.5.3, and 14.3.5.5 will have the following format.

Page 1 of X Table 14.3.5.1 Clinical Laboratory Summary and Change from Baseline - Serum Chemistry (Safety Population)

| | | | | | Trea | tment | | Ch | ange Fro | m Baseli | ne |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Laboratory Test (unit) | Normal Range# | Time<br>Point | Statistic | Α | В | C | D | Α | В | С | D |
| Parameter1 (unit) | xx - xx | Baseline* | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | <simil<br>previ</simil<br> | ar to<br>ous columns> | | lated fo | | |
| | | Day 3 | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | | | | | | |
| | | Day 6 | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | | | | | | |

<Programmer note: Similar for remaining laboratory tests and time point. Sort alphabetically by lab test name.>

Note: # Lowest of the lower ranges and highest of the higher ranges are used. Refer to Appendix 16.1.10.1 for the breakdown.

Baseline\* is Day -1 of Period 1 and Day 11 of previous period for Periods 2, 3, 4 and is the last non-missing predose measurement prior to dosing, including rechecks and unscheduled assessments. Day 11 measurement of Periods 1, 2, 3 was replicated as postdose value of Periods 1, 2, 3 and baseline value of Periods 2, 3, 4.

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >

Program: /CAXXXXX/sas prq/stsas/tab PROGRAMNAME.sas DDMMYYYYY HH:MM

## Tables 14.3.5.2, 14.3.5.4, and 14.3.5.6 will have the following format.


Table 14.3.5.2 Clinical Laboratory Shift from Baseline - Serum Chemistry (Safety Population)

| | | | Baseline L<br><br>Postdose | | Bas | Baseline N | | | Baseline H | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Tabasas | W | m' | | | e | Postdose | | se | Postdose | | |
| Laboratory<br>Test (units) | Treat-<br>ment | Time<br>Point | L | N | Н | L | N | Н | <br>L | N | Н |
| Testname(unit) | А | Day 3<br>Day 6 | X<br>X | XX | X<br>X | X<br>X | XX<br>XX | X<br>X | X<br>X | XX<br>XX | X<br>X |
| | В | Day 11<br>Day 3 | X | XX | X<br>X | X | XX | X<br>X | X | XX | X |
| | | Day 6<br>Day 11 | X<br>X | XX<br>XX | X<br>X | X<br>X | XX<br>XX | X<br>X | X<br>X | XX<br>XX | X<br>X |

<Programmer note: Similar for remaining treatments and laboratory tests. Use N = Within Normal Range, O = Outside Normal Range for urinalysis shift table.>

Note: N = Within Normal Range, L = Below Normal Range, H = Above Normal Range.

Baseline is Day -1 of Period 1 and Day 11 of previous period for Periods 2, 3, 4 and is the last non-missing predose measurement prior to dosing, including rechecks and unscheduled assessments. Day 11 measurement of Periods 1, 2, 3 was replicated as postdose value of Periods 1, 2, 3 and baseline value of Periods 2, 3, 4.

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >

Program: /CAXXXXX/sas\_prg/stsas/tab\_programname.sas DDMMMYYYY HH:MM


Table 14.3.5.7 Vital Sign Summary and Change From Baseline (Safety Population)

| 77' 1 - 3 - 0' | m' | | | Tr | reatmen | t | C | hange From | m Baseline | ) |
|---|---|---|---|---|---|---|---|---|---|---|
| Vital Sign<br>Parameter (unit) | Time<br>Point | Statistic | A | В | С | D | A | В | С | D |
| Parameter1 (unit) | Baseline* | n | XX | XX | XX | XX | | | | |
| | | Mean | XX.XX | XX.XX | XX.XX | XX.XX | | | | |
| | | SD | X.XXX | X.XXX | X.XXX | X.XXX | | | | |
| | | Minimum | XX.X | XX.X | XX.X | XX.X | | | | |
| | | Median | XX.XX | XX.XX | XX.XX | XX.XX | | | | |
| | | Maximum | XX.X | XX.X | XX.X | XX.X | | | | |
| | Hour 0.75 | n | XX | XX | XX | XX | XX | XX | XX | XX |
| | | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | SD | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
| | | Minimum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Maximum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Hour 2 | n | XX | XX | XX | XX | XX | XX | XX | XX |
| | | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | SD | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
| | | Minimum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | | Median | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | | Maximum | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

<Programmer note: Similar for remaining vital sign time points and parameters>

Note: Baseline\* is the last non-missing predose measurement prior to dosing, including rechecks and unscheduled assessments.

Treatment A: < >

Treatment B: < >

Treatment C: < >

Treatment D: < >

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Page 1 of X Table 14.3.5.8 12-Lead Electrocardiogram Summary and Change from Baseline (Safety Population)

| ROG | | Tr | reatmen | t | Change From Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| ECG<br>Parameter (unit) | Time<br>Point | Statistic | А | В | С | D | A | В | С | D |
| Parameterl (unit) | Baseline | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XXX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.X | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.X | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | | | | |
| | Hour 2 | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.X | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX |
| | Hour 4 | n<br>Mean<br>SD<br>Minimum<br>Median<br>Maximum | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.X | XX<br>XX.XX<br>X.XXX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX<br>XX.XX | XX<br>XX.XX<br>X.XX<br>XX.X<br>XX.XX<br>XX.XX |

<Programmer note: Similar for remaining time points and parameters.>

Note: Baseline\* is the last non-missing predose measurement prior to dosing, including rechecks and unscheduled assessments.

Treatment A: < >

Treatment B: < >

Treatment C: < >

Treatment D: < >

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DDMMMYYYY HH:MM

#### 11. LISTING SHELLS

The following listing shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the listings that will be presented and included in the final CSR. These listings will be generated off of the Celerion SDTM Tabulation Model 1.4 mapped in accordance with SDTM Implementation Guide 3.2. All listings will be presented in Courier New size font 9.

Actual treatment sequence will be used unless the column header uses the reference randomized sequence. Period Day will be used unless there is a footnote describing that the day referenced is using Period 1 Day 1 (ie, AE listing).


Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

| Laboratory Group | Test Name | Sex | Age Category | Reference F | Range Unit |
|---|---|---|---|---|---|
| Serum Chemistry | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| Hematology | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |
| | Test Name | XXXXXX | XX | XX - XX | units |

<Programmer note: Sort alphabetically by lab test name within each lab group.>

<similar for remaining Laboratory Groups and Test Names>


Appendix 16.2.1 Subject Discontinuation (Safety Population)

| Subject<br>Number | Randomized<br>Treatment<br>Sequence | | | . Date | Completed<br>Study? | Primary Discontinua | tion Reason |
|---|---|---|---|---|---|---|---|
| XXX-XXX | XXXX | XXXX | Post | DDMMYYYY | YES | <pre><programming note:<="" pre=""></programming></pre> | Include Specify after :> |
| XXX-XXX | XXXX | XXXX | Post | DDMMMYYYY | YES | | |
| XXX-XXX | XXXX | XXXX | Post | DDMMYYYYY | YES | | |
| XXX-XXX | XXXX | XXXX | Post | DDMMYYYYY | YES | | |
| XXX-XXX | XXXX | XX | Post | DDMMYYYY | NO | Adverse Event | |
| XXX-XXX | XXXX | XXXX | Post | DDMMYYYY | YES | | |

Note: Treatment A: < >
Treatment B: < >
Treatment C: < >

Treatment D: < >

Appendix 16.2.2 Protocol Deviations (Safety Population)


| Subject<br>Number | | | Date | Day | Assessment | Deviation<br>Type | SOP or<br>Protocol<br>Deviation | Deviation | Deviation<br>Category | |
|---|---|---|---|---|---|---|---|---|---|---|
| 001-001 | X | X | 23FEB2019 | X | | STUDY ASSESSMENTS/<br>PROCEDURES | CELERION SOP<br>GSOP.03.0011 | THE STUDY SPECIFIC "DOSING COMPLIANCE" OVERLAY (SOURCE DOCUMENTATION UTILIZED TO DOCUMENT THAT THE SUBJECT WAS INSTRUCTED NOT TO CRUSH, SPLIT, OR CHEW THE STUDY DRUG PER PROTOCOL AND THAT SUBJECTS' HANDS WERE VERIFIED TO ENSURE THAT THE STUDY DRUGS WERE INGESTED) WAS NOT COMPLETED AT THE 168.00 HOUR TIMEPOINT. | MINOR | NO ACTION/<br>FOLLOW-UP<br>REQUIRED |
| | | | 25FEB2019 | X | 8 HOUR POST<br>DOSE PK SAMPLE | LABORATORY<br>ASSESSMENTS/<br>PROCEDURE | CELERION SOP<br>GSOP.03.0040 | BLOOD COLLECTION CONDITIONS OVERLAY (SOURCE DOCUMENTATION USED BY THE COLLECTION ASSOCIATE TO DOCUMENT THAT SAMPLES WERE HANDLED ACCORDING TO THE SPECIFICATION SHEET [SOURCE DOCUMENT CONTAINING DETAILED INSTRUCTIONS FOR STUDY PROCEDURES BASED ON THE PROTOCOL]) WAS NOT COMPLETED IN ERROR. | MINOR | NO ACTION/<br>FOLLOW-UP<br>REQUIRED |

Note: Treatment A: < >

Treatment B: < >

Treatment C: < >

Treatment D: < >

Program: /CA26434/sas\_prg/stsas/lis/SDTM-LIS-DV.SAS 15MAY2019 11:29


Appendix 16.2.4.1 Demographics (Safety Population)

| Subject<br>Number | Date of<br>Birth | Age*<br>(yrs) | Sex | Race | Ethnicity | Height<br>(cm) | Weight<br>(kg) | Body Mass<br>Index<br>(kg/m^2) | Informed<br>Consent<br>Date | Informed<br>Consent<br>Version Date |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | DDMMYYYY | XX | AAAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DDMMYYYY | DDMMYYYY |
| XXX-XXX | DDMMYYYYY | XX | AAAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DDMMYYYYY | DDMMYYYYY |
| XXX-XXX | DDMMYYYYY | XX | AAAAAA | AAAAAAA | AAAAAAAAA | XXX | XX.XX | XX.XX | DDMMYYYY | DDMMYYYY |

Note: \* Age is calculated form the date of first dosing.


Appendix 16.2.4.2 Updated Informed Consent (Safety Population)

| Subject<br>Number | Date Subject Signed<br>Informed Re-Consent | Informed Re-Consent<br>Version Date | Reason for<br>Re-Consent |
|---|---|---|---|
| XXX-XXX | DDMMYYYY | DDMMYYYY | XXXXXXXXXXXX |
| XXX-XXX | DDMMYYYY | DDMMYYYY | XXXXXXXXXXXX |
| XXX-XXX | DDMMYYYY | DD <b>MM</b> YYYY | XXXXXXXXXXXX |
| XXX-XXX | DD <b>MM</b> YYYY | DDMMYYYYY | XXXXXXXXXXXXX |


#### Appendix 16.2.4.3 Physical Examination (Safety Population)

| _ | Treatment<br>Sequence | Period | Day Hour | Date | Body<br>System | Answer or<br>Result | Comment |
|---|---|---|---|---|---|---|---|
| XXX-XXX | AB | Screen | | DDMMYYYY | Was PE performed?<br>General<br>HEENT<br>< > | Yes<br>Normal<br>Normal<br>< > | |
| | | 1 | 1 -0.75 | DDMMYYYY | Was PE performed?<br>HEENT<br>< > | Yes<br>Unchanged<br>< > | |

Note: Treatment A: < >

Treatment B: < >

Treatment C: < >

Treatment D: < >


Appendix 16.2.4.4 Medical and Surgical History (Safety Population)

| | | | | | Date | | | |
|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Any<br>History? | Study<br>Period | Category | Body system | Start | End | Ongoing? | Condition or Events |
| XXX-XXX | XXX | Screen | Medical<br>Surgical | XXXXXXXXX | DDMMYYYY<br>DDMMYYYY | DDMMYYYY<br>DDMMYYYYY | YES | XXXXXXX XXXXXXX XXXXXXXX |
| XXX-XXX | XXX | Screen | Medical | XXXXXXXXXX | DDMMYYYY | DDMMYYYY | NO | |


#### Appendix 16.2.4.5 Nicotine Use (Safety Population)

| Subject<br>Number | - | Substance | Description of Use | Start<br>Date | End<br>Date |
|---|---|---|---|---|---|
| XXX-XXX | Screen | XXXXXXXX XXX | XXXXX XXXXXXX XXXXXX | DDMMYYYY | DDMMYYYY |


#### Appendix 16.2.5.1.1 Inclusion Criteria

- 1. Healthy, adult, male or female (of non-childbearing potential only), 18-55 years of age, inclusive, at screening.
- 2. <>
- 3. <>
- 4. <>
- 5. <>

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18032

Celerion, Clinical Study Report No. CA25494


#### Appendix 16.2.5.1.2 Exclusion Criteria

- 1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
- 2. <>
- 3. <>
- 4. <>
- 5. < >
- 6. <>
- 7. <>


Appendix 16.2.5.2 Subject Eligibility (Safety Population)

| Subject<br>Number | Study<br>Period | Did subject meet all eligibility criteria? | Specify |
|---|---|---|---|
| XXX-XXX | Screen | YES | |
| XXX-XXX | Screen | NO | <pre><this column="" data="" if="" is="" only="" present="" presented=""></this></pre> |


Appendix 16.2.5.3.1 Check-in Criteria

- 1. Did the Subject report any study restriction violations since the last study visit?
- 2. IF YES TO ANY QUESTION, WAS SUBJECT APPROVED FOR STUDY?

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18032

# Celerion, Clinical Study Report No. CA25494


#### Appendix 16.2.5.3.2 Check-in Responses (Safety Population)

| Subject Tre | eatment | t Study | | Check-in Criteria | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Number Sec | | | Day | Hour | Date | Time | X | X | Specify |
| XXX-XXX AE | 3 | 1 | Х | Check-in | DDMMYYYY | hh:mm | YES | YES | <pre><this column="" data="" if="" is="" only="" present="" prints=""></this></pre> |

Note: Treatment A: < >

Treatment B: < >

Treatment C: < >

Treatment D: < >
# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18032

#### Celerion, Clinical Study Report No. CA25494


#### Appendix 16.2.5.4.1 Test Compound Description

| Treatment | Compound | Form | Route |
|-----------|--------------|------|-------|
| A | XXXXXXXXXXXX | < > | XXXX |
| В | XXXXXXXXXXX | < > | XXXX |

<similar for Treatments C and D>

Programmer Note: Compound Name should be the actual compound (EXTRT) and dosage (EXTDOSE) administered (ie, per SDTM EX)

Note: Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >

## Loxo Oncology, Inc. LOXO-292, LOXO-RET-18032 Celerion, Clinical Study Report No. CA25494


Appendix 16.2.5.4.2 Test Compound Administration Times (Safety Population)

| Subject<br>Number | | Treatment | Day | Hour | Start<br>Date | Start<br>Time | Compound | Dosage | Comments |
|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | 1<br>2 | X<br>X | X<br>X | | DDMMYYYY<br>DDMMYYYY | | XXXXXXXXX | < ><br>< > | <pre><only are<br="" if="" populate="" there="">comments present in the data&gt;</only></pre> |

Note: Treatment A: < >
Treatment B: < >
Treatment C: < >

Treatment D: < >

Programmer Note: Compound Name should be the actual compound (EXTRT) administered (ie, per SDTM EX)


Appendix 16.2.5.5 PK Blood Draw Times (Safety Population)

| Subject<br>Number | _ | Treatment | Day | Hour | Date | Actual<br>Time | Bioassay | Comments |
|---|---|---|---|---|---|---|---|---|
| XXX-XXX | 1 | Χ | 1 | -X.XX | DDMMYYYY | X:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DDMMYYYYY | X:XX:XX | XXXXXXXXX | |
| | | | | XX.XX | DDMMYYYYY | X:XX:XX | XXXXXXXXX | |
| | | | | XX.XX | DDMMYYYYY | XX:XX:XX | XXXXXXXXX | |
| | | | | XX.XX | DDMMYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DDMMYYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | 2 | XX.XX | DD <b>MM</b> YYYY | X:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DDMMYYYYY | X:XX:XX | XXXXXXXXXX | |
| | | | | XX.XX | DDMMYYYYY | XX:XX:XX | XXXXXXXXXX | |
| | | | 3 | XX.XX | DDMMYYYYY | X:XX:XX | XXXXXXXXXXX | |

Note: Treatment A: < >
Treatment B: < >
Treatment C: < >

Treatment D: < >


Appendix 16.2.5.6 Meal Times (Safety Population)

| Subject<br>Number | _ | Treatment | Day | Hour | Event | Date | Start<br>Time | Stop<br>Time | Comments |
|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | 1 | A | X | -XX.XX | LUNCH | DDMMYYYY | XX:XX:XX | XX:XX:XX | |
| | | | | -XX.XX | DINNER | DDMMYYYYY | XX:XX:XX | XX:XX:XX | |
| | | | | -XX.XX | SNACK | DDMMYYYYY | XX:XX:XX | XX:XX:XX | |
| | | | X | XX.XX | LUNCH | DDMMYYYYY | XX:XX:XX | XX:XX:XX | |
| | | | | -XX.XX | DINNER | DDMMYYYYY | XX:XX:XX | XX:XX:XX | |
| | | | | -XX.XX | SNACK | DDMMYYYYY | XX:XX:XX | XX:XX:XX | |
| | | | X | XX.XX | BREAKFAST | DDMMYYYYY | XX:XX:XX | XX:XX:XX | |
| | | | | -XX.XX | LUNCH | DDMMYYYYY | XX:XX:XX | XX:XX:XX | |
| | | | | -XX.XX | DINNER | DD <b>MM</b> YYYY | XX:XX:XX | XX:XX:XX | |
| | 2 | В | -X | -XX.XX | LUNCH | DD <b>MM</b> YYYY | XX:XX:XX | XX:XX:XX | |
| | | | | -XX.XX | DINNER | DD <b>MM</b> YYYY | XX:XX:XX | XX:XX:XX | |
| | | | | -XX.XX | SNACK | DD <b>MM</b> YYYY | XX:XX:XX | XX:XX:XX | |
| | | | X | XX.XX | BREAKFAST | DDMMYYYY | XX:XX:XX | XX:XX:XX | |
| | | | | XX.XX | LUNCH | DDMMYYYY | XX:XX:XX | XX:XX:XX | |
| | | | | XX.XX | DINNER | DDMMYYYY | XX:XX:XX | XX:XX:XX | |
| | | | | -XX.XX | SNACK | DDMMYYYYY | XX:XX:XX | XX:XX:XX | |
| | | | X | XX.XX | BREAKFAST | DDMMYYYY | XX:XX:XX | XX:XX:XX | |
| | | | | -XX.XX | LUNCH | DDMMYYYYY | XX:XX:XX | XX:XX:XX | |
| | | | | -XX.XX | DINNER | DDMMYYYYY | XX:XX:XX | XX:XX:XX | |

Note: Treatment A: <>

Treatment B: < >

Treatment C: < >

Treatment D: < >

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18032

#### Celerion, Clinical Study Report No. CA25494


#### Appendix 16.2.5.7 Prior and Concomitant Medications (Safety Population)

| Subject Treat-<br>Number ment | _ | | Medication<br>(WHO* Term) | Dosage | Route | Frequency | Start<br>Day/Date/Time | Stop<br>Day/Date/Time | | | Continuing Medication? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX<br>XXX-XXX X | No<br>Yes | Yes | None<br>ACETAMINOPHEN<br>(ACETAMINOPHEN | | BY MOUTH | AS NEEDED | XX/DDMMMYYYY/<br>HH:MM | XX/DDMMYYYY/<br>HH:MM | XXXXX | XXX | YES |

Note:  $\star$  Concomitant medications are coded with WHO Dictionary Version 01-Mar-2019 b3.

^ Med = Medication; UNK = Unknown

Prior medication was medication taken prior to study drug administration.

Start and stop day is relative to Period 1 Day 1.

Treatment A: < >

Treatment B: < >

Treatment C: < >

 ${\tt Treatment D:} \; < \; > \;$ 


#### Appendix 16.2.7.1 Adverse Events (I of II) (Safety Population)

| | | | | Time from<br>Last Dose | | Onset | | | Resolved | | Duration |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Treatment | TE?^ | Adverse Event/<br>Preferred Term* | (DD:HH:MM) | Day | Date | Time | Day | Date | Time | (DD:HH:MM) |
| XXX-XXX | | None | | | | | | | | | |
| XXX-XXX | X | Yes | XXXXXXXXXXXX/<br>XXXXXXXXXX | XX:XX:XX | XX | DDMMYYYY | X:XX | XX | DDMMYYYY | X:XX | XX:XX:XX |
| | | No | XXXXXXXXXXXXX/<br>XXXXXXXXXX | XX:XX:XX | XX | DDMMYYYY | X:XX | XX | DDMMYYYY | X:XX | XX:XX:XX |

Note: \* Adverse events are classified according to MedDRA Version 22.0 by System Organ Class and Preferred Term.

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >

<sup>^</sup> TE = Treatment-emergent, Onset and resolved day is relative to Period 1 Day 1.

## Loxo Oncology, Inc. LOXO-292, LOXO-RET-18032 Celerion, Clinical Study Report No. CA25494


#### Appendix 16.2.7.2 Adverse Events (II of II) (Safety Population)

| | | 7.1 | | Onset | | | | | | Act | ion for | Other | Relatio | onship to |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>Number | Treat-<br>ment | - Adverse<br>Event | Day | Date | Time | Freq^ | Severity | Ser* | Outcome | LOXO-292 | Moxifloxacin | Action<br>Taken | LOXO-292 | Moxifloxacin |
| XXX-XXX | | None | | | | | | | | | | | | |
| XXX-XXX | Х | XXXXXXX | XX | DDMMYYYY | XX:XX | Inter. | Grade 1 | NO | Resolved | Dose Not<br>Changed | Dose Not<br>Changed | None | | Not Related to Moxifloxacin |

Note: Ser\* = Serious; Freq^ represents Frequency: SI = Single Episode, Inter. = Intermittent, Cont. = Continuous Severity/Intensity: Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe or medically significant but not immediately life-threatening; Grade 4 = Life-threatening consequences; Grade 5 = Death related to AE

Not all grades are appropriate for all AEs, therefore some AEs are listed in the CTCAE with fewer than 5 options for grade selection.

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18032

## Celerion, Clinical Study Report No. CA25494


#### Appendix 16.2.7.3 Adverse Event Non-Drug Therapy (Safety Population)

| | | | Onset | | | Resolved | | Therapy | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject Ad | | Adverse | | | | | | | | | |
| Number | 2 | | Day | Date | Time | Day | Date | Time | Date | Time | Description |
| XXX-XXX | X | DRY LTPS | XX | DDMMYYYY | X:XX | XX | DDMMYYYY | X:XX | DDMMMYYYY | XX:XX | PETROLEUM JELLY |

Note: Onset and resolved day is relative to Period 1 Day 1.

Treatment A: < >
Treatment B: < >

Treatment C: < >

 ${\tt Treatment D:} \; < \; > \;$ 

# Loxo Oncology, Inc. LOXO-292, LOXO-RET-18032

## Celerion, Clinical Study Report No. CA25494


#### Appendix 16.2.7.4 Adverse Event Preferred Term Classification (Safety Population)

| | | | | | | Onset | |
|---|---|---|---|---|---|---|---|
| Subject | | Adverse | | | | | |
| Number | Treatment | Event | Preferred Term* | Body System | Day | Date | Time |
| XXX-XXX | X | XXXXXXX XXXXX XXXX XXXXXX | XXXXXXXXX XXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XX | DDMMYYYYY | X:XX |

Note: \* Adverse events are classified to MedDRA Version 22.0 by System Organ Class and Preferred Term.

Onset day is relative to Period 1 Day 1.

Treatment A: < >

Treatment B: < >
Treatment C: < >

Treatment D: < >

#### Appendices 16.2.8.1.2-16.2.8.1.4 will have the following format.


Appendix 16.2.8.1.1 Clinical Laboratory Report - Serum Chemistry (Safety Population)

| Subject<br>Number | _ | reatment<br>equence | Study<br>Period | Day | Hour | Date | Parameter1<br>< Range><br>(Unit) | Parameter2<br>< Range><br>(Unit) | Parameter3<br>< Range><br>(Unit) | Parameter4<br>< Range><br>(Unit) | Parameter5<br>< Range><br>(Unit) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XX/M | XXXX | Screen<br>1<br>2 | -X<br>X<br>X<br>X | CHECK-IN<br>X<br>X<br>X | DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY<br>DDMMMYYYY | XX HN<br>XX<br>XX<br>XX<br>XX LY- | XX LN XX XX XX | XX<br>XX<br>XX<br>XX<br>XX | XX XX LY- | XX HN<br>XX<br>XX<br>XX<br>XX<br>XX |

Programmer Note: Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for. Arrange alphabetically by lab test name.

Add fourth flag in the cases that ^ or R are used for the PI flag. This flag will be found in the ClinQuick Extraction

Note: \$ Age is calculated from the date of first dosing.

H = Above Reference Range, L = Below Reference Range
Computer Clinical Significance: N = Not Clinically Significant, Y = Clinically Significant
PI Interpretation: - = Not Clinically Significant, R = To be Rechecked, ^ = Will be Retested at a Later Event
Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >

## Loxo Oncology, Inc. LOXO-292, LOXO-RET-18032 Celerion, Clinical Study Report No. CA25494


#### Appendix 16.2.8.1.5 Clinical Laboratory Report - Comments (Safety Population)

| _ | Treatment<br>Sequence | | Day | Hour | Date | Department | Test | Result | Unit | Comment |
|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | XXXX | X | X | -X.X | DDMMYYYY | Other Tests | Fibrinogen | XXX | ٥. | Not significant in the context of this study. |


Appendix 16.2.8.2 Vital Signs (Safety Population)

| 0.1. | Q1 1 | | | | | | Blood P | ressur | re (mmHg) | D 1 | - | Temper- | ** ' 1 ' | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| _ | Study<br>Period | | | Hour | Date | Time | Position | Arm | Sys/Dia | Pulse<br>(bpm) | ation<br>(rpm) | ature<br>(°C) | Weight<br>(kg) | Comments |
| XXX-XXX | Screen | | | | DDMMYYYY | X:XX:XX | | | | | | | XXX.X | |
| | | | | | DDMMYYYYY | X:XX:XX | SUPX | Right | XXX/ XX | XX | XX | XX.X | | |
| | X | X | -X | Check-in | DDMMYYYYY | XX:XX:XX | | | | | | | XXX.X | |
| | | | | | DDMMYYYYY | XX:XX:XX | SUPX | Right | XXX/ XX | XX | XX | | | |
| | | | X | X.X | DD <b>MM</b> YYYY | XX:XX:XX | SUPX | Right | • | | | | | |
| | | | | X.X | DDMMYYYYY | XX:XX:XX | SUPX | Right | | | | | | |
| | | | | X.X | DDMMYYYYY | X:XX:XX | SUPX | Right | XXX/ XX | XX | XX | | | |
| | | | | X.X | DDMMYYYY | X:XX:XX | SUPX | Right | XXX/ XX | XX | XX | | | |
| | | | | X.X | DDMMYYYY | X:XX:XX | SUPX | Right | XXX/ XX | XX | XX | | | |
| | | | | R | DD <b>MM</b> YYYY | XX:XX:XX | SUPX | Right | XXX/ XX | XX | XX | | | |
| | | | | X.X | DDMMYYYY | XX:XX:XX | SUPX | Right | | | | | | |

Programmer note: Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for.

Note: SUPX = X-minute supine, R = Recheck Value, Sys/Dia = Systolic/Diastolic, rpm = breaths per minute

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >


Appendix 16.2.8.3 12-Lead Electrocardiogram (Safety Population)

| Subject<br>Number | Study<br>Period | Treatment | Day | Hour | Date | Time | Result | Heart<br>Rate<br>(bpm) | PR<br>(msec) | QRS<br>(msec) | QT<br>(msec) | QTcF*<br>(msec) | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| XXX-XXX | Screen | | | | DDMMYYYY | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | 1 | X | -1 | Check-in | DDMMYYYYY | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | | | | X.XX | DDMMYYYYY | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | 2 | X | X | X.XX | DDMMYYYYY | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | | | | X.XX | DDMMYYYYY | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X | |
| | | | X | X.XX | DDMMYYYYY | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X # | |
| | | | X | ^ X.XX | DDMMYYYYY | X:XX:XX | NORMAL | XX | XXX.X | XX.X | XXX.X | XXX.X @ | |

Programmer note: Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for.

Note: NCS = Abnormal, Not Clinically Significant

QTcF\* = QT corrected for heart rate using Fridericia's correction.

# = QTcF > 450, @ = QTcF change from baseline greater than 30 msec

^ = Repeat assessment or unscheduled event

Treatment A: < >

Treatment B: < >
Treatment C: < >

Treatment D: < >

## Loxo Oncology, Inc. LOXO-292, LOXO-RET-18032 Celerion, Clinical Study Report No. CA25494


Appendix 16.2.8.4 Holter Monitoring Times (Safety Population)

| Subject | Study | | St<br> | art<br> | | | Stop<br> | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Number | _ | Day | Hour | Date | Time | Day | Hour | Date | Time | Comment |
| XXX-XXX | X | X | XX.XX | DDMONYYYY | XX:XX | X | XX.XX | DDMONYYYY | XX:XX | <pre><only if="" populated="" present=""></only></pre> |

## Loxo Oncology, Inc. LOXO-292, LOXO-RET-18032 Celerion, Clinical Study Report No. CA25494


#### Appendix 16.2.8.5 Phone Call (Safety Population)

| Subject<br>Number | Study<br>Period | Day | Phone Call Completed? | Date | Time | If no, reason |
|---|---|---|---|---|---|---|
| XXX-XXX | X | X | Yes/No | DDMMYYYY | HH:MM | Wrong number |



# Statistical Analysis Plan

# A Single-Dose, Randomized, Double-Blind, Placebo- and Positive-Controlled, 4-Way Crossover Study to Evaluate the Effect of LOXO-292 on the QTc Interval in Healthy Adult Subjects

**Protocol: LOXO-RET-18032** 

Sponsor: Loxo Oncology, Inc.

**ERT Internal ID: 266-1001** 

**Version:** Final 1.0

**Authors:** PPD , MS, Biostatistician I

PPD , PhD, Senior Biostatistician

**Date:** 22 July 2019



# **Revision History**

| Version | Issue Date | Author(s) | Description |
|---|---|---|---|
| Draft 0.1 | 23 May 2019 | PPD and | Initial version for review. |
| | | PPD | |
| Draft 0.2 | 17 June 2019 | PPD and | Revised version. |
| | | PPD | |
| Draft 0.3 | 10 July 2019 | PPD | Revised version to add testing for carryover effect. |
| Draft 0.4 | 19 July 2019 | PPD | Revised version. |
| Final 1.0 | 22 July 2019 | PPD | Final version. |



## **Table of Contents**

| 1 | Abbreviations | 4 |
|---|---------------------------------------------------------------|----|
| 2 | Introduction | 5 |
| 3 | Study Design | 5 |
| 4 | Cardiodynamic ECG Assessment | 5 |
| | 4.1 Cardiodynamic ECG Objectives | 6 |
| | 4.1.1 Primary Objective | |
| | 4.1.2 Secondary Objectives | |
| | CCI | |
| | 4.2 Cardiodynamic ECG Endpoints | 7 |
| | 4.2.1 Primary Endpoint | 7 |
| | 4.2.2 Secondary Endpoints | 7 |
| | CCI | |
| 5 | Statistical Methods | 7 |
| | 5.1 General Methodology | 7 |
| | 5.2 Analysis Populations | 9 |
| | 5.3 Baseline | 9 |
| | 5.4 QT Correction Methods | |
| 6 | Analyses | |
| | 6.1 Carryover Effect Test | |
| | 6.2 Concentration-QTc Analysis (Analysis of Primary Endpoint) | |
| | 6.2.1 Investigation of Hysteresis | |
| | 6.2.2 Appropriateness of a Linear Model | |
| | 6.3 Assay Sensitivity | |
| | 6.4 Categorical Analysis | |
| | 6.5 By-Time Point Analysis | |
| | 6.6 Determination of Sample Size | |
| 7 | References | |
| 8 | Tables, Figures, and Listings | |
| | 8.1 Tables | |
| | 8.2 Figures | |
| | 8.3 Listings | 19 |
| Q | Approvals | 20 |



# 1 Abbreviations

| Abbreviation | Term/Description |
|------------------|--------------------------------------------------|
| bpm | Beats per minute |
| CI | Confidence interval |
| C <sub>max</sub> | Maximum plasma concentration |
| C-QT | Concentration-QTc |
| Δ | Change-from-baseline |
| ΔΔ | Placebo-corrected change-from-baseline |
| ECG | Electrocardiogram |
| HR | Heart rate |
| LOESS | Locally weighted scatter plot smoothing |
| LS | Least squares |
| ms | Millisecond |
| PK | Pharmacokinetic(s) |
| PR | PR interval of the ECG |
| Q-Q | Quantile-quantile |
| QRS | QRS interval of the ECG |
| QT | QT interval of the ECG |
| QTc | Corrected QT interval |
| QTcF | Corrected QT interval using Fridericia's formula |
| QTcP | Population heart rate-corrected QT interval |
| RR | RR interval of the ECG |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SE | Standard error |
| TQT | Thorough QT |



#### 2 Introduction

This statistical analysis plan (SAP) was developed after review of the protocol LOXO-RET-18032 (Final version dated 03 April 2019) for the study "A Single-Dose, Randomized, Double-Blind, Placebo-and Positive-Controlled, 4-Way Crossover Study to Evaluate the Effect of LOXO-292 on the QTc Interval in Healthy Adult Subjects" and the ERT contract/proposal. This document defines the populations to be analyzed and provides full details of the statistical analyses, data displays, and algorithms to be used for data derivations to aid in the production of the statistical output and the statistical section of the cardiac safety report in regard to electrocardiogram (ECG) and concentration-QTc analyses. Relevant subject characteristics as well as the electrocardiographic parameters that will be evaluated are described along with the specific statistical methods.

## 3 Study Design

This is a single-dose, randomized, double-blind (except for the use of moxifloxacin), placebo- and positive-controlled, 4-way crossover study. Thirty-two, healthy, adult male and female (women of non-childbearing potential only) subjects will be enrolled.

Screening of subjects will occur within 28 days prior to the first dosing. On Day 1, subjects will be randomized to 1 of 4 treatment sequences.

On Day 1 of each period, subject will receive 1 of 2 single oral dose levels of LOXO-292, a single oral dose of moxifloxacin, or a single oral dose of LOXO-292 matching placebo on 1 occasion, according to a randomization scheme. Cardiodynamic samples will be collected pre-dose and for up to 24 hours post-dose as outlined below. Pharmacokinetic (PK) samples will be collected pre-dose and for up to 24 hours post-dose for moxifloxacin and up to 240 hours post-dose for LOXO-292, as per treatment received. There will be a washout period of 10 days between dosing in each period.

Safety and tolerability will be assessed through end of treatment or early termination by monitoring adverse events, performing physical examinations and clinical laboratory tests, measuring vital signs, and recording ECGs.

## 4 Cardiodynamic ECG Assessment

Holter monitors will be used to collect continuous 12-lead ECG data for the purpose of collecting cardiodynamic ECGs for approximately 26 hours. Recording will be started and stopped at logistically optimal times to ensure that all scheduled time points are collected. At least three 12-lead ECG recordings will be extracted from the Holter monitor data on Day 1 of each period within a 5-minute time window around the scheduled time points, but prior to the PK blood sample collection.

The time points for ECG extraction in each period are 0.75, 0.5, and 0.25 hours prior to dosing on Day 1 and 0.25, 0.5, 0.75, 1.5, 2, 2.5, 3, 4, 7, 9, 12, and 24 hours post-dose (the 24 hours post-dose time point will occur on Day 2, at the end of the Day 1 Holter recording).



Timing and recording technique for ECGs will be standardized for all subjects. Subjects will be required to lie quietly in a supine position with minimal movement and minimal exposure to noise and other environmental stimuli (e.g., TV, loud radio, interactions with other participants, etc.) for at least 10 minutes before and 5 minutes during the ECG extraction to allow for quality ECG extraction. All ECG extraction should occur in a 5-minute time window around the scheduled/nominal time. If targeted ECG time points are artefactual or of poor quality, analyzable 10-second ECGs will be extracted as close as possible to the targeted time points.

Nominal time of the ECG recording will be used for the cardiodynamic analyses.

All Holter/ECG data will be collected using M12R continuous 12-lead digital recorders and the M12A Enterprise Holter System Client (Global Instrumentation, LLC, Manlius, New York, USA). The equipment will be supplied and supported by ERT.

ECG intervals will be measured by the core laboratory in a blinded manner using the Expert Precision QT technique (see Appendix A for more details). The ECG database will be locked before any statistical analysis is undertaken.

#### 4.1 Cardiodynamic ECG Objectives

For the purpose of this analysis plan, objectives related to ECG assessment are described.

#### 4.1.1 Primary Objective

The primary ECG objective is to evaluate the effects of therapeutic and supratherapeutic exposure of LOXO-292 on the QTc interval by assessing concentration-QT relationship using exposure-response modelling.

#### 4.1.2 Secondary Objectives

- To assess the effect of therapeutic and supratherapeutic exposure of LOXO-292 on other ECG parameters (heart rate [HR], PR, and QRS interval);
- To demonstrate sensitivity of this QTc assay using moxifloxacin as a positive control in healthy adult subjects;
- To assess the effect of therapeutic and supratherapeutic exposure of LOXO-292 on categorical outliers for HR, PR, and QRS interval.





## 4.2 Cardiodynamic ECG Endpoints

#### 4.2.1 Primary Endpoint

The primary endpoint is the effect of LOXO-292 plasma concentrations on the QTc interval using linear mixed-effect exposure-response modeling, including the predicted  $\Delta\Delta$ QTc at C<sub>max</sub> values corresponding to exposure levels of interest.

#### 4.2.2 Secondary Endpoints

The secondary endpoints are:

- The change in other ECG parameters such as QT, PR, and RR intervals, QRS duration, and HR.
- Morphological changes of ECG waveform (e.g., T-wave morphology and presence of pathologic U wave).
- Determination of assay sensitivity using exposure-response modeling of the ΔΔQTc following moxifloxacin administration.



#### 5 Statistical Methods

## 5.1 General Methodology

All statistical analyses will be performed using the statistical software SAS for Windows Version 9.4 or higher (SAS Institute, Inc., Cary, NC). In all calculations, zero will be substituted for concentrations below the quantification limit of the assay and for concentrations from subjects who received placebo. Data collected from all randomized subjects will be presented in data listings. Both absolute values and change-from-baseline values for each subject will be given where applicable. All continuous data will be listed with the same precision as will be presented in the database. Data listings will be sorted by treatment, subject ID, and time point. Missing values will be represented by an empty cell and no imputation will be made.

Continuous data will be summarized using descriptive statistics including number of subjects (n), mean, median, standard deviation (SD), standard error (SE), 90% confidence interval (CI), minimum, and maximum by treatment and time point. Mean and median values will be rounded to the nearest tenth, or to the first non-zero decimal. SD, SE, and CI will be rounded to the nearest hundredth, or to 1 digit more than the nearest non-zero digit. For the concentration-QTc analysis, 3 significant digits will be kept for the effect estimates. *P* values will be reported with 4 digits and *P* values less than 0.0001 will be reported as < 0.0001. Categorical data will be summarized 2 ways, by subject and by time point. Subject data will be summarized using the count of distinct subjects that fall into the category and the percentage of the total number of subjects. Time point data will be summarized using the count of time points at which the assessments fall into the category and the percentage of the total number of time points at



which assessments are performed. Percentages will be rounded up or down to the nearest tenths decimal place. Counts (either number of subjects or number of time points) for each treatment will be used as the denominator in the calculation of percentages unless otherwise specified.



#### 5.2 Analysis Populations

The analysis populations for cardiodynamic ECG assessment are defined as follows (Table 1).

Table 1 Analysis populations for cardiodynamic ECG assessment

| Population | Subjects |
|---|---|
| Safety population | All subjects enrolled in the study who receive at least 1 dose of study drug (LOXO-292, moxifloxacin, or placebo). |
| PK population | All subjects who receive a dose of LOXO-292 or moxifloxacin and have at least 1 evaluable PK plasma concentration of LOXO-292 or moxifloxacin. |
| Cardiodynamic population | All subjects in the Safety population with measurements at baseline as well as on-treatment with at least 1 post-dose time point with a valid $\Delta QTcF$ value. The Cardiodynamic population will be used for the by-time point and categorical analyses of the cardiodynamic ECG parameters. |
| C-QT population | All subjects who are in both the PK and Cardiodynamic populations with at least 1 pair of post-dose PK and QTcF data from the same time point as well as subjects in the Cardiodynamic population who received placebo. The C-QT population will be used for the concentration-QTc analysis. This population will be defined separately for LOXO-292 and for moxifloxacin. |

#### 5.3 Baseline

For all continuous ECG parameters from each period, baseline is defined as the average of the measured ECG intervals from the 3 pre-dose time points (0.75, 0.5, and 0.25 hours before dosing) on Day 1 for the respective period.

## 5.4 QT Correction Methods

The QT and RR value for each beat will be used for HR correction. Replicate ECGs will be extracted in up to 10 replicates from each nominal time point prespecified in the protocol. The median value from each extracted replicate from evaluable beats will be calculated, and then the average of all available medians (minimum 3 medians) from a nominal time point will be used as the subject's reportable value at that time point.

The Fridericia's correction QTcF is defined as QTcF =  $QT/RR^{1/3}$ .

In case a substantial heart rate effect (i.e., largest mean  $\Delta\Delta$ HR > 10 bpm) is observed, additional QT correction methods, including the population heart rate-corrected QT interval (QTcP as described by Tornøe et al<sup>1</sup>), will be considered.



# 6 Analyses

#### 6.1 Carryover Effect Test

Before the concentration-QTc analysis in Section 6.2 is performed, it is necessary to test the carryover effect, even the possibility that some subjects receiving placebo may have small residual exposures to LOXO-292 present. A mixed-effect repeated measures model will be considered with ΔQTcF as the dependent variable; period, time (i.e., post-dose time points), treatment (therapeutic dose of LOXO-292, supratherapeutic dose of LOXO-292, and placebo), time-by-treatment interaction, period-by-treatment interaction, period-by-time interaction, and period-by-treatment-by-time as fixed effects, and baseline QTcF as a covariate. An unstructured covariance matrix will be specified for the repeated measures at post-dose time points for subject within treatment period. If the model with an unstructured covariance matrix fails to converge, other covariance matrices such as compound symmetry and autoregressive will be considered. The model will also include a subject-specific random effect. If the period-by-treatment interaction (and period-by-treatment-by-time interaction if necessary) is not statistically significant at the significance level 5%, this indicates that there is no carryover effect. Then the proposed concentration-QTc analysis (as well as by-time point analysis and categorical analysis) will be performed, and zero will be substituted for concentrations below the quantification limit of the assay and for concentrations from subjects who received placebo. Otherwise, a sensitivity analysis(es) of concentration-QTc, by-time point, and categorical analyses will be performed by excluding period(s) with observed non-zero concentrations at baseline for subjects receiving placebo. Additional sensitivity analyses may exclude subjects with more than extremely low LOXO-292 concentrations.

## 6.2 Concentration-QTc Analysis (Analysis of Primary Endpoint)

The concentration-QTc analysis will be based on the C-QT population. The relationship between LOXO-292 plasma concentration and change-from-baseline QTcF ( $\Delta$ QTcF) will be quantified using a linear mixed-effects model with  $\Delta$ QTcF as the dependent variable, LOXO-292 plasma concentration as the explanatory variate (0 for placebo), centered baseline QTcF (i.e., baseline QTcF for individual subject subtracting the population mean baseline QTcF for all subjects in the same period) as an additional covariate, study treatment (active = 1 or placebo = 0), and time (i.e., post-dose time point) as categorical factors, and a random intercept and slope per subject (Garnett et al²). The degrees of freedom for the model estimates will be determined by the Kenward-Roger method. From the model, the slope (i.e., the regression parameter for the concentration) and the treatment effect-specific intercept (defined as the difference between active and placebo) will be estimated together with the 2-sided 90% CI. The estimates for the time effect will be reported with degrees of freedom and SE.

The geometric mean of the individual  $C_{max}$  values for LOXO-292 plasma concentrations for subjects in each of the LOXO-292 dose groups will be determined, respectively. The predicted effect and its 2-sided 90% CI for  $\Delta\Delta QTcF$  (i.e., slope estimate × concentration + treatment effect-specific intercept) at this geometric mean  $C_{max}$  will be obtained. If the upper bound of the 2-sided 90% CI of the model-predicted QTc effect is below 20 ms at clinically relevant plasma levels of LOXO-292, it will be concluded that LOXO-292 does not cause clinically concerning QTc prolongation within the observed plasma concentration ranges.



The plot of the observed median-quantile LOXO-292 concentrations and associated mean placeboadjusted  $\Delta QTcF$  (i.e.,  $\Delta \Delta QTcF$ ) with 90% CI adjusted for diurnal effects, together with the regression line presenting the predicted  $\Delta \Delta QTcF$  (90% CI) (as described by Tornøe et al¹) will be used to evaluate the adequacy of the model fit to the assumption of linearity and the impact on quantifying the concentration-QTc relationship. The observed  $\Delta QTcF$  values from the active groups will be adjusted by the estimated time effect from the concentration-QTc model (i.e. the estimated diurnal effect under the placebo treatment). The individually estimated placebo-adjusted  $\Delta QTcF_{i,j}$  equals the individual  $\Delta QTcF_{i,j}$  for subject i administered with LOXO-292 at time point j minus the estimation of time at time point j (i.e., time effect). Additional plots will be used to validate the model assumptions. For evaluation of the heart rate-corrected QT interval, a scatter plot and quantile plot of QTcF and RR intervals by treatment with a regression line and a linear mixed-effects line (90% CI), respectively, will also be given. Exploratory analyses (via graphical displays and/or model fitting) will also include accounting for a delayed effect (hysteresis) and the justification for the choice of pharmacodynamics model (linear versus nonlinear).

The SAS code for the concentration-QTc analysis is as follows:

```
PROC MIXED DATA=PKPD method=reml;
CLASS SUBJID TIME;
MODEL DQTC=TRT CONC TIME CBASE/ solution cl noint alpha=0.1 alphap=0.1 COVB DDFM=KR;
RANDOM INT CONC /type=UN SUBJECT=SUBJID s;
ESTIMATE 'Pred Mean Diff for T1' TRT 1 CONC &GeoMeanCmax_1 / CL ALPHA=0.1;
ESTIMATE 'Pred Mean Diff for T2' TRT 1 CONC &GeoMeanCmax_2 / CL ALPHA=0.1;
RUN;
```

Where PKPD=C-QT population, SUBJID=subject number, TRT=treatment (active=1 or placebo=0), TIME=nominal time point, CONC=plasma concentration of LOXO-292, CBASE=centered baseline QTcF, T1= therapeutic dose of LOXO-292, T2 = supratherapeutic dose of LOXO-292, GeoMeanCmax\_1=geometric mean  $C_{max}$  for therapeutic dose of LOXO-292, GeoMeanCmax\_2=geometric mean  $C_{max}$  for supratherapeutic dose of LOXO-292, and DQTC= $\Delta$ QTcF.

#### 6.2.1 Investigation of Hysteresis

Hysteresis will be assessed based on joint graphical displays of the least squares (LS) mean difference between  $\Delta QTcF$  under LOXO-292 and under placebo ( $\Delta\Delta QTcF$ ) for each post-dose time point from the by-time point analysis and the mean concentration of LOXO-292 at the same time points. In addition, hysteresis plots will be given for LS mean  $\Delta\Delta QTcF$  from the by-time point analysis and the mean concentrations. If a QT effect > 20 ms (i.e., LS mean  $\Delta\Delta QTcF > 10$  ms) cannot be excluded and the mean peak  $\Delta QTcF$  effect is observed at the same time point and the delay between peak plasma levels and peak QT effect of more than 1 hour is present, other concentration-QTc models such as a model with an effect compartment may be explored. With the provision stated above, hysteresis will be assumed if the curve of hysteresis plot shows a counterclockwise loop. A significant treatment effect-specific intercept is not biologically plausible and therefore may be indicative of hysteresis, if it cannot be explained by a nonlinear relationship.



#### 6.2.2 Appropriateness of a Linear Model

To assess the appropriateness of a linear model, normal Q-Q plots for the standardized residuals and the random effects, and plots of standardized residuals versus concentration, fitted values, centered baseline QTcF, nominal time, and active treatment will be produced. Scatter plots for standard residuals versus continuous covariates and box plots for standard residuals versus discrete covariates will be provided. The scatter plots of standardized residuals versus concentration, and centered baseline QTcF by LOESS fitting (i.e., locally weighted scatter plot smoothing (as described by Cleveland³) will also be produced with optimal smoothing parameters selected by the Akaike information criterion with a correction. A scatter plot of observed concentration and  $\Delta$ QTcF with a LOESS smooth line with 90% CI and a linear regression line will also be provided to check the assumption of a linear concentration-QTc relationship. If there is an indication that a linear model is inappropriate, additional models will be fitted, in particular an  $E_{max}$  model. The concentration-QTc analysis will then be repeated for the model found to best accommodate the nonlinearity detected.

#### 6.3 Assay Sensitivity

The analysis to show assay sensitivity will be based on the concentration-QTc analysis of the effect on  $\Delta QTcF$  of goal moxifloxacin using a similar model as for the primary analysis. That is, the relationship between moxifloxacin plasma concentration and  $\Delta QTcF$  will be investigated by linear mixed-effects modeling. The model will include  $\Delta QTcF$  as the dependent variable, moxifloxacin plasma concentration as the explanatory variate (0 for placebo), centered baseline QTcF as an additional covariate, study treatment (moxifloxacin = 1 or placebo = 0), and time (i.e., post-dose time point) as categorical factors, and a random intercept and slope per subject (Garnett et al<sup>1</sup>). The geometric mean of the individual  $C_{max}$  values for subjects receiving the single dose of graph moxifloxacin will be determined. The predicted effect and its 2-sided 90% CI for  $\Delta\Delta QTcF$  (i.e., slope estimate × concentration + treatment effect-specific intercept) at this geometric mean  $C_{max}$  will be obtained.

If the slope of the moxifloxacin plasma concentration/ $\Delta$ QTcF relationship is statistically significant at the 10% level in a 2-sided test and the lower bound of the 2-sided 90% CI of the predicted QT effect at the observed geometric  $C_{max}$  of the column dose is above 5 ms, assay sensitivity will be deemed to have been demonstrated.

## 6.4 Categorical Analysis

Results for categorical outliers, T-wave morphology, and U-wave presence will be summarized in frequency tables with counts and percentages for both number of subjects and number of time points.

A subject or time point will be determined as an outlier if the following criteria (which are assessed separately) are met for the ECG intervals (Table 2). Each subject meeting a categorical threshold will be counted once, using the largest value.



Table 2 Criteria for determining a subject or time point outlier

| ECG<br>interval | Categorical outlier criteria |
|---|---|
| QTcF | Treatment-emergent value of $>$ 450 and $\le$ 480 ms when not present at baseline (new onset) |
| | Treatment-emergent value of > 480 and ≤ 500 ms when not present at baseline (new onset) |
| | Treatment-emergent value of > 500 ms when not present at baseline (new onset) |
| | Increase of QTcF from baseline of > 30 and ≤ 60 ms |
| | Increase of QTcF from baseline > 60 ms |
| PR | Increase of PR from baseline > 25% resulting in PR > 200 ms |
| QRS | Increase of QRS from baseline > 25% resulting in QRS > 120 ms |
| HR | Decrease of HR from baseline >25% resulting in HR < 50 bpm |
| | Increase of HR from baseline >25% resulting in HR > 100 bpm |

All outliers will be summarized for each treatment on the basis of incidence rates. A subject will be counted only once for a particular outlier event if the subject experiences more than 1 episode of that event. The total number of time points will be based on the number of observed time points across all subjects within a treatment group.

For T-wave morphology and U-wave presence, treatment-emergent changes will be assessed, i.e., changes not present at baseline. For each category of T-wave morphology and of U-waves, the category will be deemed as present if observed in all replicates at the time point. For baseline, the category will be deemed as present if observed in any replicates from all time points that constitute baseline, i.e., the 3 time points prior to dosing on Day 1 in each period.

The T-wave morphology and U-wave presence categories are described as follows (Table 3).

Table 3 T-wave morphology and U-wave presence categories (assessed manually)

| Category | Description |
|---|---|
| Normal T-wave (+) | Any positive T-wave not meeting any criterion below. |
| Flat T-wave | T-amplitude < 1 mm (either positive or negative), including flat isoelectric line. |
| Notched T-wave (+) | Presence of notch(es) of at least 0.05 mV amplitude on ascending or descending arm of the positive T-wave. |
| Biphasic | T-wave that contains a second component with an opposite phase that is at least 0.1 mV deep (both positive/negative and negative/positive and polyphasic T-waves included). |



| Category | Description |
|---|---|
| Normal T-wave (-) | T-amplitude is negative, without biphasic T-wave or notches. |
| Notched T-wave (-) | Presence of notch(es) of at least 0.05 mV amplitude on descending or ascending arm of the negative T-wave. |
| U-waves | Presence of abnormal U-waves. |

#### 6.5 By-Time Point Analysis

The "by time point analysis" will be based on cardiodynamic population. The "by time point analysis" for QTcF will be based on a mixed-effect repeated measures model with ΔQTcF as the dependent variable; period, time (i.e., post-dose time point: categorical), treatment (therapeutic dose of LOXO-292, supratherapeutic dose of LOXO-292, moxifloxacin, and placebo), and time-by-treatment interaction as fixed effects; and baseline QTcF as a covariate. An unstructured covariance matrix will be specified for the repeated measures at post-dose time points for subject within treatment period. If the model with an unstructured covariance matrix fails to converge, other covariance matrices such as compound symmetry and autoregressive will be considered. The model will also include a subject-specific random effect. If the fixed effect for period should prove to be not significant (i.e., if the *P* value > 0.1), the fixed effect may be removed from the model and the analysis will be repeated without period. From this analysis, the LS mean and 2-sided 90% CI will be calculated for the contrast "LOXO-292 versus placebo" at each dose of LOXO-292 and each post-dose time point, separately. If a carry-over effect is observed (Section 6.1), the period-by-treatment interaction and the period-by-treatment-by-time interaction will also be included in the model.

For HR, PR, and QRS intervals, the analysis will be based on the post-dose  $\Delta$ HR,  $\Delta$ PR, and  $\Delta$ QRS. The same (by-time point analysis) model will be used as described for QTcF. The LS mean, SE, and 2-sided 90% CI from the statistical modeling for both change-from-baseline and placebo-corrected change-from-baseline values will be listed in the tables and graphically displayed.

The SAS code for the by-time point analysis for QTcF is as follows:

PROC MIXED DATA=ECG; CLASS SUBJID TREAT TIME PERIOD SEQUENCE; MODEL DQTC=BASE TREAT TIME TREAT\*TIME PERIOD SEQUENCE/DDFM=KR; random intercept / SUBJECT = SUBJID type=UN; REPEATED TIME / SUBJECT = SUBJID\*PERIOD type = un; LSMEANS TREAT\*TIME/CL DIFF ALPHA=0.1; RUN;

Where ECG=Cardiodynamic population, SUBJID=subject identifier, TREAT=treatment (therapeutic dose of LOXO-292, supratherapeutic dose of LOXO-292, moxifloxacin, and placebo), TIME=nominal time point, BASE= baseline QTcF, PERIOD=period, SEQUENCE=sequence, and DQTC=ΔQTcF.



## 6.6 Determination of Sample Size

The sample size determination is based on testing to support a non-inferiority hypothesis, with a non-inferiority margin of 10 ms for this determination. Using non-inferiority margin of 10 ms, assuming a 1-sided 0.05 significance level and a common within-subject SD of 8 ms for QTc, a sample size of 30 evaluable subjects (allowing for 2 dropouts) would be expected to provide at least  $\frac{100}{300}$ % power to detect an expected mean difference of 3 ms in  $\Delta$ QTc between LOXO-292 and placebo.

The proposed 4-way crossover design in this study, using 32 subjects randomized to 1 of 4 treatment sequences will result in up to 32 sets of observations each for moxifloxacin and placebo. Given what was reported in the literature, this sample size is deemed appropriate to detect a drug-induced QTc prolongation by moxifloxacin of greater than 5 ms.



#### 7 References

- 1. Tornøe CW, Garnett CE, Wang Y, Florian J, Li M, Gobburu JV. Creation of a knowledge management system for QT analyses. *J Clin Pharmacol*. 2011;51(7):1035-1042.
- 2. Garnett C, Bonate PL, Dang Q, Ferber G, Huang D, Liu J, et al. Scientific white paper on concentration-QTc modeling. [Published correction appears in *J Pharmacokinet Pharmacodyn*. 2018;45(3):399]. *J Pharmacokinet Pharmacodyn*. 2018;45(3):383-397.
- 3. Cleveland WS. Robust locally weighted regression and smoothing scatterplots. *J Am Stat Assoc.* 1979;74(368):829-836.
- 4. Hurvich CM, Simonoff JS, and Tsai CL. Smoothing parameter selection in nonparametric regression using an improved Akaike Information Criterion. *J R Stat Soc Series B Stat Methodol*. 1998;60(2):271-293.

## 8 Tables, Figures, and Listings

#### 8.1 Tables

| Number | Title | Comments |
|---|---|---|
| 14.2.3.1.1 | Baseline values of ECG parameters with descriptive statistics | Number of subjects (n), mean, SD, SE, 90% CI, median, minimum, and maximum from descriptive analysis will be given by treatment for each ECG parameter. |
| 14.2.3.1.2 | Absolute values of ECG parameters with descriptive statistics | n, mean, SD, SE, 90% CI, median, minimum, and maximum from descriptive statistics will be given by treatment and post-dose time point for each ECG parameter. |
| 14.2.3.1.3.1-<br>14.2.3.1.3.2 | Change-from-baseline QTcF, HR, PR, and QRS (ΔQTcF, ΔHR, ΔPR, and ΔQRS) at each time point | n, LS mean, SE, and 90% CI from the statistical modeling will be given by treatment and time point (Section 6.5). |
| 14.2.3.1.4.1-<br>14.2.3.1.4.4 | Placebo-corrected change-from-<br>baseline QTcF, HR, PR, and QRS<br>( $\Delta\Delta$ QTcF, $\Delta\Delta$ HR, $\Delta\Delta$ PR, and<br>$\Delta\Delta$ QRS) at each time point | LS mean, SE, and 90% CI from the statistical modeling will be given by treatment and time point (Section 6.5). |
| 14.2.3.1.5 | QTcF outliers per absolute category across treatment groups | Number (%) of subjects and time points with QTcF > $450$ and $\le 480$ ms, $> 480$ and $\le 500$ ms, and $> 500$ ms by treatment (Section 6.4). |
| 14.2.3.1.6 | QTcF outliers per change-from-<br>baseline category across treatment<br>groups | Number (%) of subjects and time points with $\Delta QTcF > 30$ and $\leq 60$ ms, and $> 60$ ms by treatment (Section 6.4). |



| Number | Title | Comments |
|---|---|---|
| 14.2.3.1.7 | Categorical analysis for HR, PR, and QRS groups | Number (%) of subjects and time points with $\Delta PR > 25\%$ and $PR > 200$ ms at post-baseline; $\Delta QRS > 25\%$ and $QRS > 120$ ms at post-baseline; $PR = 100$ HR decrease from baseline $PR = 100$ by at post-baseline; and $PR = 100$ by at post-baseline (Section 6.4). |
| 14.2.3.1.8 | T-wave morphology and U-wave presence across treatment: treatment-emergent changes across treatment groups | Number (%) of subjects and time points falling into each of T-wave categories: Normal (+), Flat, Notched (+), Biphasic, Normal (-), Notched (-) as defined in Section 6.4. |
| 14.2.3.1.9.1 | Concentration-QTc analysis of LOXO-292 and associated ΔQTcF prolongation | Fixed-effect estimations and corresponding $P$ values will be given (Section 6.2). |
| 14.2.3.1.9.2 | Assay sensitivity analysis of moxifloxacin and associated ΔQTcF prolongation | Fixed-effect estimations and corresponding $P$ values will be given (Section 6.3). |
| 14.2.3.1.10.1 | Predicted ΔΔQTcF interval at geometric mean peak LOXO-292 concentration | Section 6.2. |
| 14.2.3.1.10.2 | Predicted ΔΔQTcF interval at geometric mean peak moxifloxacin concentration | Section 6.3. |

# 8.2 Figures

| Number | Title | Comments |
|---|---|---|
| 14.2.3.2.1 | Absolute QTcF across time points | Mean and 90% CI from descriptive analysis will be given by treatment. |
| 14.2.3.2.2.1-<br>14.2.3.2.2.4 | Change-from-baseline QTcF, HR, PR, and QRS ( $\Delta$ QTcF, $\Delta$ HR, $\Delta$ PR, and $\Delta$ QRS) across time points | LS mean and 90% CI from the statistical modeling will be shown by treatment for each parameter (Section 6.5). |
| 14.2.3.2.3.1-<br>14.2.3.2.3.4 | Placebo-corrected change-from-<br>baseline QTcF, HR, PR, and QRS<br>( $\Delta\Delta$ QTcF, $\Delta\Delta$ HR, $\Delta\Delta$ PR, and<br>$\Delta\Delta$ QRS) across time points | LS mean and 90% CI from the statistical modeling will be shown by treatment (Section 6.5). |
| 14.2.3.2.4.1 | Scatter plot of QTcF versus RR by treatment | Scatter plots of QTcF and RR intervals by treatment with regression lines will be given (Section 6.2). |
| 14.2.3.2.4.2 | QTcF-RR quantile plot by treatment | QTcF-RR quantile plots (with quantiles) with linear mixed-effects line and 90% CI will be given (Section 6.2). |
| 14.2.3.2.5.1 | Plot of mean LOXO-292 plasma concentrations over time | Section 6.2. |



| Number | Title | Comments |
|---|---|---|
| 14.2.3.2.5.2 | Plot of mean moxifloxacin plasma concentrations over time | Section 6.3. |
| 14.2.3.2.6 | Joint plot of LOXO-292 plasma concentrations and $\Delta\Delta QTcF$ over time | Section 6.2.1. |
| 14.2.3.2.7 | Hysteresis plot of LOXO-292 plasma concentration and $\Delta\Delta QTcF$ connected in temporal order | This is what is often called a "Hysteresis plot" (Section 6.2.1). |
| 14.2.3.2.8.1 | Scatter plot of observed LOXO-292 plasma concentrations and ΔQTcF by subject | Scatter plot of $\Delta QTcF$ versus concentration with LOESS line and 90% CI and simple linear regression line (Section 6.2). |
| 14.2.3.2.8.2 | Scatter plot of observed LOXO-292 plasma concentrations and estimated placebo-adjusted $\Delta QTcF$ by subject | Scatter plot of estimated placebo-adjusted $\Delta QTcF$ versus observed concentration and linear mixed-effect regression line with CI (Section 6.2). |
| 14.2.3.2.8.3 | Scatter plot of observed moxifloxacin plasma concentrations and ΔQTcF by subject | Scatter plot of $\Delta QTcF$ versus concentration with LOESS line and 90% CI and simple linear regression line (Section 6.3). |
| 14.2.3.2.8.4 | Scatter plot of observed moxifloxacin plasma concentrations and estimated placebo-adjusted $\Delta QTcF$ by subject | Scatter plot of estimated placebo-adjusted $\Delta QTcF$ versus concentration and linear mixed-effect regression line with CI (Section 6.3). |
| 14.2.3.2.9.1 | Model-predicted ΔΔQTcF (mean and 90% CI) and estimated placeboadjusted ΔQTcF (mean and 90% CI) across deciles of LOXO-292 plasma concentrations | Section 6.2. |
| 14.2.3.2.9.2 | Model-predicted ΔΔQTcF (mean and 90% CI) and estimated placeboadjusted ΔQTcF (mean and 90% CI) across deciles of moxifloxacin plasma concentrations | Section 6.3. |
| 14.2.3.2.10.1 | Predicted ΔΔQTcF interval at geometric mean peak LOXO-292 concentrations | Section 6.2. |
| 14.2.3.2.10.2 | Predicted ΔΔQTcF interval at geometric mean peak moxifloxacin concentrations | Section 6.3. |
| 14.2.3.2.11.1 | Scatter plot of standardized residuals versus fitted values for LOXO-292 | Section 6.2.2. |
| 14.2.3.2.11.2 | Scatter plot of standardized residuals versus fitted values for moxifloxacin | Section 6.3. |



| Number | Title | Comments |
|---|---|---|
| 14.2.3.2.12.1 | Scatter plot of standardized residuals versus LOXO-292 concentrations with LOESS | Section 6.2.2. |
| 14.2.3.2.12.2 | Scatter plot of standardized residuals versus moxifloxacin concentrations with LOESS | Section 6.3. |
| 14.2.3.2.13.1 | Scatter plot of standardized residuals versus centered baseline QTcF with LOESS for LOXO-292 | Section 6.2.2. |
| 14.2.3.2.13.2 | Scatter plot of standardized residuals versus centered baseline QTcF with LOESS for moxifloxacin | Section 6.3. |
| 14.2.3.2.14.1 | Box plot of standardized residuals versus nominal time for LOXO-292 | Section 6.2.2. |
| 14.2.3.2.14.2 | Box plot of standardized residuals versus nominal time for moxifloxacin | Section 6.3. |
| 14.2.3.2.15.1 | Box plot of standardized residuals versus treatment for LOXO-292 | Section 6.2.2. |
| 14.2.3.2.15.2 | Box plot of standardized residuals versus treatment for moxifloxacin | Section 6.3. |
| 14.2.3.2.16.1 | Normal Q-Q plot of standardized residuals for LOXO-292 | Section 6.2.2. |
| 14.2.3.2.16.2 | Normal Q-Q plot of standardized residuals for moxifloxacin | Section 6.3. |
| 14.2.3.2.17.1 | Normal Q-Q plots of the estimated random effects for LOXO-292 | Section 6.2.2. |
| 14.2.3.2.17.2 | Normal Q-Q plots of the estimated random effects for moxifloxacin | Section 6.3. |

# 8.3 Listings

| Number | Title | Comments |
|---|---|---|
| 16.2.6.3.1<br>-<br>16.2.6.3.4 | QTcF, HR, PR, and QRS parameters – absolute and change-from-baseline values | Section 6.5. |
| 16.2.6.4 | T-wave morphology and U-wave presence | Section 6.4. |
| 16.2.6.5 | ΔQTcF and time-matched concentrations of LOXO-292 and moxifloxacin for each subject | Data for concentration-QTc (Section 6.2) and assay sensitivity (Section 6.3). |



## 9 Approvals



Chief Scientific Officer, Cardiac Safety





Project Manager



22 JUL 2019





24-Jul-19 | 18:15:46 PDT -

Date

Statistical Analysis Plan for Loxo Oncology, Inc. Study LOXO-RET-18032 Final Version 1.0

Page 20 of 21 CONFIDENTIAL



## **Appendix A: Expert Precision QT Analysis**

Expert Precision QT analysis (formerly High Precision QT analysis) will be performed on all analyzable (non-artifact) beats in the 10 ECG replicates (1 replicate consists of one 14 second ECG). Statistical quality control procedures will be used to review and assess all beats and identify "high" and "low" confidence beats using several criteria including:

- QT or QTc values exceeding or below certain thresholds (biologically unlikely)
- RR values exceeding or below certain thresholds (biologically unlikely)
- Rapid changes in QT, QTc, or RR from beat to beat

Placement of fiducials and measurements of all primary ECG parameters (QT, QTc, RR) in all recorded beats of all replicates will be performed using the iCOMPAS software. All beats that are deemed "high confidence" will not be reviewed by an ERT ECG analyst. All low confidence beats will be reviewed manually by an ERT ECG analyst and adjudicated using pass-fail criteria. The beats found acceptable by manual review will be included in the analysis. The beats confirmed to meet fail criteria will not be included in the analysis.

For the purpose of measuring PR and QRS intervals and to assess T-wave morphology and presence of U-waves, the TQT Plus algorithm will select the 3 ECG replicates with the highest quality score from the ECG extraction window. These 3 ECGs will be analyzed using a semi-automated process to determine these parameters. If 3 consecutive usable beats cannot be identified in at least 2 of the 3 replicates, then all beats in all replicates will be reviewed for that time point using a manual analysis.

If manual analysis is required, then all beats in a minimum of 3 replicates will be reviewed using the iCOMPAS software. The ERT ECG analyst will review all usable beats in Lead II (or an alternate lead) for each replicate and will review and/or adjust the fiducial placements (onset of P, onset of Q, offset of S, and offset of T-wave that were electronically marked) of each waveform and also document the T-wave morphology and the presence of U-waves for each beat. A replicate will only be reported if it has 3 approved, usable beats.